### CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN for

DMID Protocol: 17-0010 Study Title:

A Phase 2A Partially-blind Placebo Controlled Trial to Evaluate the Safety and Immunogenicity of Live Attenuated, Intranasal *B. pertussis* vaccine (BPZE1) in Healthy Adults

NCT03541499

Version 1.0

DATE: 29-OCT-2019

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

#### **STUDY TITLE**

A Phase 2A Partially-blind Placebo Controlled Trial to Evaluate the Safety and Immunogenicity of Live Attenuated, Intranasal B. pertussis vaccine (BPZE1) in Healthy Adults

| <b>Protocol Number Code:</b> | DMID Protocol: 17-0010 |
|---|---|
| <b>Development Phase:</b> | Phase 2a |
| Products: | One dose (10 <sup>7</sup> CFU or 10 <sup>9</sup> CFU) of lyophilized, live-attenuated <i>Bordetella pertussis</i> vaccine (BPZE1) manufactured by |
| Form/Route: | Intranasal |
| Indication Studied: | B. pertussis |
| Sponsor: | Division of Microbiology and Infectious Diseases National Institute of Allergy and Infectious Diseases National Institutes of Health |
| Clinical Trial Initiation Date: | 14SEP2018 |
| Clinical Trial Completion Date: | 15MAY2020 |
| Date of the Analysis Plan: | 29OCT2019 |
| Version Number: | 1.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

### TABLE OF CONTENTS

| STUDY T | TITLE | II |
|---|---|---|
| TABLE O | F CONTENTS | III |
| LIST OF A | ABBREVIATIONS | VI |
| 1. | PREFACE | 1 |
| 2. | INTRODUCTION | 2 |
| 2.1. | Purpose of the Analyses | 3 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 4 |
| 3.1. | Study Objectives | 4 |
| 3.1.1. | Primary Objective | 4 |
| 3.1.2. | Secondary Objectives | 4 |
| 3.2. | Endpoints | 4 |
| 3.2.1. | Primary Outcome Measures | 4 |
| 3.2.2. | Secondary Outcome Measures | 4 |
| 3.3. | Study Definitions and Derived Variables | 5 |
| 4. | INVESTIGATIONAL PLAN | 6 |
| 4.1. | Overall Study Design and Plan | 6 |
| 4.2. | Discussion of Study Design, Including the Choice of Control Groups | |
| 4.3. | Selection of Study Population | 6 |
| 4.4. | Treatments | 6 |
| 4.4.1. | Treatments Administered | 6 |
| 4.4.2. | Identity of Investigational Product(s) | 6 |
| 4.4.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 6 |
| 4.4.4. | Selection of Doses in the Study | 7 |
| 4.4.5. | Selection and Timing of Dose for Each Subject | 7 |
| 4.4.6. | Blinding | 7 |
| 4.4.7. | Prior and Concomitant Therapy | 7 |
| 4.4.8. | Treatment Compliance | 8 |
| 4.5. | Efficacy (Immunogenicity) and Safety Variables | 8 |
| 4.5.1. | Safety Variables | 8 |
| 4.5.2. | Immunogenicity Variables | 8 |
| 4.5.3. | Nasal Clearance Variables | 8 |

### **Table of Contents** (continued)

| 5. | SAMPLE SIZE CONSIDERATIONS | 9 |
|---|---|---|
| 6. | GENERAL STATISTICAL CONSIDERATIONS | 10 |
| 6.1. | General Principles | 10 |
| 6.2. | Timing of Analyses | 10 |
| 6.3. | Analysis Populations | 10 |
| 6.3.1. | Safety Population | 10 |
| 6.3.2. | Immunogenicity Population. | 10 |
| 6.3.3. | Per Protocol Population | 10 |
| 6.4. | Covariates and Subgroups | 11 |
| 6.5. | Missing Data | 11 |
| 6.6. | Interim Analyses and Data Monitoring | 11 |
| 6.6.1. | Interim Safety Review | 11 |
| 6.6.2. | Interim Immunogenicity Review | 12 |
| 6.7. | Multicenter Studies | 12 |
| 6.8. | Multiple Comparisons/Multiplicity | 12 |
| 7. | STUDY SUBJECTS | 13 |
| 7.1. | Disposition of Subjects | 13 |
| 7.2. | Protocol Deviations | 13 |
| 8. | EFFICACY EVALUATION | 14 |
| 8.1. | Secondary Immunogenicity Analysis | 14 |
| 9. | SAFETY EVALUATION | 15 |
| 9.1. | Demographic and Other Baseline Characteristics | 15 |
| 9.1.1. | Prior and Concurrent Medical Conditions | 15 |
| 9.1.2. | Prior and Concomitant Medications | 15 |
| 9.2. | Measurements of Treatment Compliance | 15 |
| 9.3. | Adverse Events | 15 |
| 9.3.1. | Solicited Events and Symptoms | 16 |
| 9.3.2. | Unsolicited Adverse Events | 16 |
| 9.4. | Deaths, Serious Adverse Events and other Significant Adverse Events | 16 |
| 9.5. | Pregnancies | 17 |
| 9.6. | Clinical Laboratory Evaluations | 17 |
| 9.7. | Vital Signs and Physical Evaluations | 17 |

### **Table of Contents** (continued)

| 9.8. | Concomitant Medications | 17 |
|--------|---------------------------------------------------------|-----|
| 9.9. | Other Safety Measures | 18 |
| 10. | PHARMACOKINETICS | 19 |
| 11. | IMMUNOGENICITY | 20 |
| 12. | OTHER ANALYSES | 21 |
| 13. | REPORTING CONVENTIONS | 22 |
| 14. | TECHNICAL DETAILS | 23 |
| 15. | SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY ANALYSES | |
| 16. | REFERENCES | 25 |
| 17. | LISTING OF TABLES, FIGURES, AND LISTINGS | 26 |
| APPEND | ICES | 27 |
| APPEND | IX 1. TABLE MOCK-UPS | 28 |
| APPEND | IX 2. FIGURE MOCK-UPS | 123 |
| APPEND | IX 3. LISTINGS MOCK-UPS | 135 |

### LIST OF ABBREVIATIONS

| AE | Adverse Event |
|-----------|--------------------------------------------------|
| AESI | Adverse Event of Special Interest |
| ALT | Alanine Aminotransferase |
| aPV | Acellular Pertussis Vaccine |
| BP | Blood Pressure |
| BPZE1 | Live Attenuated, Intranasal B. pertussis vaccine |
| С | Celsius |
| CFU | Colony Forming Units |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| Desc. | Description |
| dL | Deciliter |
| DMID | Division of Microbiology and Infectious Diseases |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| ELISA | Enzyme-linked Immunosorbent Assay |
| F | Fahrenheit |
| FHA | Filamentous Hemagglutinin |
| FIM | Fimbriae |
| GMT | Geometric Mean Titer |
| GMFR | Geometric Mean Fold Rise |
| Hgb | Hemoglobin |
| HIV | Human Immunodeficiency Virus |
| ICH | International Conference on Harmonisation |
| ITT | Intention to Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MedDRA PT | MedDRA Preferred Term |
| mg | Milligram |
| mL | Milliliter |
| N | Number (typically refers to subjects) |

### **List of Abbreviations** (continued)

| NIH | National Institutes of Health |
|--------|------------------------------------------|
| NOCMCs | New Onset Chronic Medical Conditions |
| PP | Per Protocol |
| PRN | Pertactin |
| PT | Pertussis Toxin |
| RCD | Reverse Cumulative Distribution |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SDCC | Statistical and Data Coordinating Center |
| SMC | Safety Monitoring Committee |
| SOC | System Organ Class |
| VUMC | Vanderbilt University Medical Center |
| U | Units |
| μL | Microliter |
| WBC | White Blood Cell |
| WHO | World Health Organization |
| wPV | Whole Cell Pertussis Vaccine |

#### 1. PREFACE

The Statistical Analysis Plan (SAP) for "A Phase 2A Partially-blind Placebo Controlled Trial to Evaluate the Safety and Immunogenicity of Live Attenuated, Intranasal *B. pertussis* vaccine (BPZE1) in Healthy Adults" (DMID Protocol 17-0010) describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures planned for the final analyses. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains a review of the study design, general statistical considerations, comprehensive statistical analysis methods for efficacy and safety outcomes, and a list of proposed tables and figures. Within the table, figure, and listing mock-ups (Appendices 1, 2, and 3), references to CSR sections are included. Any deviation from this SAP will be described and justified in the CSR, as appropriate. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

#### 2. INTRODUCTION

Bordetella pertussis (B. pertussis) is a gram-negative bacterium and a causative agent of pertussis colonizing infection, a precursor to the disease more commonly known as whooping cough. A recent publication modeling pertussis cases and deaths estimated there were 24.1 million pertussis cases and 160,700 deaths in children younger than 5 years in 2014 worldwide.[1] Despite the dramatic decline in Whooping Cough cases and deaths in industrialized nations during the 20th Century due to public health vaccine initiatives, recent decades have witnessed a sharp increase in cases.

Two types of pertussis vaccines are available worldwide: whole cell Pertussis vaccine (wPV) and acellular Pertussis vaccine (aPV). Although aPV overcomes several potential adverse effects of wPV (e.g. fever and seizures) and is the only pertussis vaccine marketed in the U.S., the protective efficacy of aPV appears to be lower than wPV with induced immunity waning in about 4-12 years. Additionally, the high cost of aPV limits its use in developing countries.

Acellular pertussis vaccines (aPVs have several deficiencies that have contributed to pertussis outbreaks across the US and around the world. Young infants are especially vulnerable but are not fully protected until they complete a 3 dose aPV vaccination series, at about 7 months of age. Preclinical baboon studies suggest that aPV does not prevent nasopharyngeal colonization and, hence, does not prevent transmission from adults and adolescents to vulnerable infants.[2] Multiple published studies in various countries have demonstrated high rates of subclinical (asymptomatic) *B. pertussis* colonizing infections. [3-6]. Mathematical models predict that asymptomatic *B. pertussis* colonization is the most probable cause of the surge in pertussis rates. [7] Thus, a need exists for an adult and adolescent vaccine that induces potent and durable systemic immunity, but also mucosal immunity to prevent nasopharyngeal colonization and transmission to infants.

Since the best-known method of inducing both potent systemic and mucosal immunity is by natural *B. pertussis* infection, BPZE1 was constructed through

Over 20 peer-reviewed publications have demonstrated the preclinical safety and efficacy of the live-attenuated vaccine [8-11], and two Phase 1 clinical studies [12, 13] have demonstrated safety and immunogenicity at various doses in healthy adults.



The main advantage of the lyophilized BPZE1 formulation over the liquid formulation is long-term stability and storage at refrigeration temperature instead of storage at very low freezing temperature. The primary purpose of this Phase 2a study is to evaluate the safety and immunogenicity of the lyophilized formulation. The hypothesis for this trial is that lyophilized BPZE1, administered intranasally, will be sufficiently safe and immunogenic.

### 2.1. Purpose of the Analyses

These analyses will assess the safety, tolerability, immunogenicity, and nasal clearance of a single intranasal dose of either 10<sup>7</sup> or 10<sup>9</sup> colony forming units (CFU) of lyophilized BPZE1 vaccine. The protocol for DMID 17-0010 calls for a planned preliminary analysis on safety, immunogenicity, and B. pertussis colonization data through Day 46 (or Day 29 if no subjects remain colonized with B. pertussis at the Day 29 visit). The preliminary report may be made available to DMID and the vaccine company partner and to the lead principal investigator for planning subsequent trials. Interim analyses will not be used to make any decisions concerning the conduct of this trial. This Statistical Analysis Plan encompasses the analyses to be included in the preliminary report and final CSR.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

### 3.1. Study Objectives

#### 3.1.1. Primary Objective

• To assess the safety and tolerability of a single intranasal dose of either 10<sup>7</sup> or 10<sup>9</sup> colony forming units (CFU) of lyophilized BPZE1 vaccine.

#### 3.1.2. Secondary Objectives

- To assess the humoral immunogenicity of lyophilized BPZE1 vaccine at Day 15, Day 29 and Day 181 following receipt of one intranasal dose of 10<sup>7</sup> or 10<sup>9</sup> CFU of BPZE1.
- To assess mucosal immunogenicity of lyophilized BPZE1 vaccine at Day 29 and Day 181 following receipt of one intranasal dose of 10<sup>7</sup> or 10<sup>9</sup> CFU of BPZE1.
- To evaluate nasal clearance of BPZE1 by culture at Day 29 (and if still positive, at Day 46) following receipt of one intranasal dose of lyophilized BPZE1 vaccine of 10<sup>7</sup> or 10<sup>9</sup> CFU of BPZE1.

### 3.2. Endpoints

#### 3.2.1. Primary Outcome Measures

- Occurrence of solicited local and systemic reactogenicity from the time of the study vaccination through 14 days post-vaccination
- Occurrence of unsolicited non-serious adverse events from the time of the study vaccination through 28 days post-vaccination
- Occurrence of serious adverse events (SAEs) and new onset chronic medical conditions (NOCMCs) from the time of the study vaccination through approximately Day 181 post vaccination
- Occurrence of adverse events of special interest through approximately Day 29 post vaccination

#### 3.2.2. Secondary Outcome Measures

#### Humoral Immune Response

- Geometric mean titers (GMTs) by serum IgG and IgA ELISA to PT, FHA, PRN, FIM 2/3 on Days 1, 15, 29, and 181
- Geometric mean fold rise (GMFR) by serum IgG and IgA ELISA to PT, FHA, PRN, FIM 2/3 on Days 15, 29 and 181 relative to baseline (Day 1)
- The proportion of subjects that achieve seroconversion (defined as ≥2-fold rise from baseline) to individual pertussis antigens (PT, FHA, PRN, and FIM 2/3) by serum IgG or IgA ELISA at Days 15, 29, 181 or any time point relative to baseline (Day 1)
- Proportion of subjects achieving seroconversion (serum IgG or IgA ELISA) to one or more pertussis antigens at Days 15, 29, 181 or any time point, relative to baseline (Day 1)

• Proportion of subjects achieving seroconversion (serum IgG/IgA ELISA) to two or more pertussis antigens at Days 15, 29, 181 or any time point, relative to baseline (Day 1)

#### Mucosal Immune Response

- Geometric mean titer ratios (GMTRs) and ratio of antigen-specific IgA ELISA (PT-IgA, FHA-IgA, PRN-IgA, FIM-IgA) to total IgA by nasal aspirate at screening, and Days 29 and 181.
- Fold rise of the ratio of antigen-specific IgA (PT-IgA, FHA-IgA, PRN-IgA, FIM-IgA) to total IgA by nasal aspirate from the screening visit to Days 29 and 181
- The proportion of subjects that achieve seroconversion (defined as ≥2-fold rise of the ratio from baseline) to individual pertussis antigens (PT, FHA, PRN, and FIM 2/3) by nasal aspirate IgA ELISA at Days 29 and 181 or any time point relative to baseline (screening)
- Proportion of subjects that achieve seroconversion (≥2-fold rise of the ratio from baseline) to at least 1 antigen (PT, FHA, PRN, or FIM 2/3) by nasal aspirate IgA ELISA from the screening visit to Days 29 and/or 181.

#### Nasal Clearance

- Proportion of subjects with detectable B. pertussis from nasopharyngeal cultures at Day 29.
- For those who remain positive at Day 29, the subjects with detectable B. pertussis at Day 46 will also be evaluated and reported. Detection of B. pertussis in culture will be assumed to be due to study-product administration.

#### 3.3. Study Definitions and Derived Variables

New Onset Chronic Medical Conditions (NOCMCs) will be defined as new medical conditions, not present at the time of screening or enrollment, that require ongoing medical care and intervention.

Achievement of seroconversion based on humoral response will be defined as a  $\geq$ 2-fold rise from baseline. Achievement of seroconversion based on mucosal response will be defined as a  $\geq$ 2-fold rise the ratio of antigen-specific IgA ELISA (PT-IgA, FHA-IgA, PRN-IgA, FIM-IgA) to total IgA by nasal aspirate from baseline.

Medically Significant Wheezing will be defined as clinician (licensed to make medical diagnoses) documented wheezing on PE accompanied by any one or more of the following: Respiratory distress (tachypnea, retractions or dyspnea), Hypoxemia (O2 saturation <95%), new prescription, or use of daily bronchodilator therapy (not on an "as needed" basis).

#### 4. INVESTIGATIONAL PLAN

#### 4.1. Overall Study Design and Plan

This is a phase 2a, single center, randomized, partially blind (i.e. the method of vaccination will be known), placebo controlled, clinical trial in which 50 healthy males and non-pregnant females 18-49 years of age who meet all eligibility criteria receive either BPZE1 10<sup>7</sup> CFU administered via VaxINator: BPZE1 10<sup>9</sup> CFU administered via VaxINator: placebo administered via VaxINator: BPZE1 10<sup>9</sup> CFU administered via Needleless Tuberculin Syringe, randomized in a 3:3:3:1 ratio. Subjects will be screened by medical history, physical exam, and clinical laboratory tests, including a urine or serum pregnancy test for women of childbearing potential. A schematic of the study design is presented in Figure 1.

#### 4.2. Discussion of Study Design, Including the Choice of Control Groups

This study is designed to obtain preliminary estimates of the safety and immune response induced by the BPZE1 lyophilized vaccine. Fifteen placebo recipients are included in order to partially blind the subjects and observer.

#### 4.3. Selection of Study Population

The study population for DMID protocol 17-0010 is males and non-pregnant females, 18 to 49 years old, inclusive, who are in good health and meet all eligibility criteria. Potential subjects will be screened from the general population at VUMC by history, physical exam, clinical laboratory tests including White Blood Cells (WBC), Hemoglobin (Hgb), platelets, serum IgG antibodies, alanine aminotransferase (ALT), Creatinine, and Human Immunodeficiency Virus (HIV), and a urine or serum pregnancy test. Potential subjects with close contact, defined as sharing a household, serving as a healthcare worker, or working professionally in settings with repeated exposures, with children less than 1 year of age or with persons with known immunocompromising conditions will be excluded. Otherwise eligible potential subjects experiencing an acute illness, including temperature >100°F, will be eligible for postponed enrollment within the screening window or rescreening once symptoms resolve.

#### 4.4. Treatments

#### 4.4.1. Treatments Administered

Subjects are administered one dose (either  $10^7$  CFU or  $10^9$  CFU) of lyophilized, live-attenuated *Bordetella pertussis* vaccine (BPZE1) or placebo.

#### 4.4.2. Identity of Investigational Product(s)

| The investigational BPZE1 ly | ophilized vaccine is for nasal administration | and contains |
|---|---|---|
| | The place | bo consists of the same constituent |
| in the same quantities as the E | SPZE1 investigational vaccines, absent the | . Both |
| were provided by | | |

#### 4.4.3. Method of Assigning Subjects to Treatment Groups (Randomization)

Enrollment/randomization will be performed through the enrollment module in the electronic data capture system, maintained by the SDCC. Eligible subjects will be randomized and assigned in a 3:3:3:1 ratio to BPZE1 10<sup>7</sup> CFU administered via VaxINator: BPZE1 10<sup>9</sup> CFU administered via VaxINator: placebo

administered via VaxINator: BPZE1 10<sup>9</sup> CFU administered via Needleless Tuberculin Syringe. The randomization is based on a block scheme to provide an approximately balanced allocation to the treatment groups during the study.

#### 4.4.4. Selection of Doses in the Study

In a Phase 1a clinical study, a dose of  $10^7$  CFU of the liquid formulation of BPZE1 administered nasally resulted in colonization of the mucosal surface in 42% of subjects with no serious adverse events. [12] In a Phase 1b clinical study, also using the liquid formulation administered nasally, but in a greater volume (400  $\mu$ L per nostril), doses of  $10^7$ ,  $10^8$ , and  $10^9$  CFU all resulted in colonization in  $\geq$ 75% of subjects with faster colonization rate and faster clearance rate being correlated with higher dosage. [13] No serious adverse events were observed in any of the dosage groups and there were no detectable differences in adverse events between dosage groups. The lyophilized formulation is hypothesized to share similar safety characteristics with the liquid formulation.

#### 4.4.5. Selection and Timing of Dose for Each Subject

Subjects are assigned randomly to treatment groups in a 3:3:3:1 ratio (BPZE1 10<sup>7</sup> CFU administered via VaxINator: BPZE1 10<sup>9</sup> CFU administered via VaxINator: placebo administered via VaxINator: BPZE1 10<sup>9</sup> CFU administered via needleless tuberculin syringe). Each subject will receive a single intranasal dose in clinic on Day 1. Timing of dose is not specified.

#### 4.4.6. Blinding

This is a partially-blind clinical trial as the method of immunization (i.e. VaxINator vs. needleless syringe) will be known. After reconstitution and transfer to a 1-mL syringe, the  $10^7$  CFU dose investigational vaccine and the placebo are transparent and indistinguishable while the  $10^9$  CFU dose can be discriminated from the placebo and the  $10^7$  CFU dose due to its opaque appearance. Therefore, syringes will be wrapped with a colored sleeve to avoid potential unblinding of study personnel or the subject. Investigators, the subject, and study personnel will remain blinded to allocation of BPZE1 or placebo.

The randomization scheme will be generated by the SDCC and provided to unblinded study personnel (i.e., research pharmacists performing study vaccination preparations and unblinded study vaccine administrators) at the participating VTEU site.

The unblinded study vaccine administrator is a study personnel member credentialed to administer vaccines and may also participate in dose preparation but will not be involved in study-related assessments or have subject contact for data collection following study vaccine administration. Laboratory personnel performing immunogenicity assays will be blinded to study assignment.

Upon request by the participating VTEU site, and at the discretion of DMID, unmasking may occur after all data have been locked at Day 181, analyzed, interpreted, and the final CSR has been completed. The Safety Monitoring Committee (SMC) may receive data in aggregate and presented by treatment arm. The SMC may also be provided with expected and observed rates of the expected AEs in an unblinded fashion and may request the treatment arm be unblinded for an individual subject if required for safety assessment. The SMC will review grouped and unblinded data in the closed session only.

#### 4.4.7. Prior and Concomitant Therapy

Administration of medications, therapies, or vaccines will be recorded on the appropriate data collection form. Concomitant medications will include all current medications and medications taken within 30 days prior to

signing the informed consent form through approximately 28 days after study vaccination (or through the early termination visit if prior to that time). Prescription and over-the-counter drugs will be included, as well as herbals, vitamins and supplements. In addition, receipt of non-study vaccines will be solicited through approximately 181 days after study vaccination and reported in the eCRF.

#### 4.4.8. Treatment Compliance

Subject compliance is not expected to be an issue because all subjects are to receive a single dose of study product administered in the clinic by a study personnel member who is unblinded to subject treatment assignment.

### 4.5. Efficacy (Immunogenicity) and Safety Variables

See Table 1 and Table 2for a schedule of study procedures.

#### 4.5.1. Safety Variables

Safety will be assessed by the frequency and severity of:

- 1. Serious adverse events (SAE) occurring from the time of vaccination through approximately 6 months after vaccination.
- 2. Solicited Adverse Events reactogenicity events occurring from the time of each study vaccination through 14 days after study vaccination:
  - **a.** Mucosal reactions including runny nose, stuffy nose/congestion, nasal pain/irritation, epistaxis, sneezing, sinus pressure/pain, sore throat, cough, and shortness of breath, cough, rhinorrhea, and sneezing
  - **b.** Systemic reactions including fever, chills, fatigue, malaise, myalgia, arthralgia, headache, and hypersensitivity.
- 3. Unsolicited Adverse Events study vaccine-related non-serious adverse events occurring from the time of study vaccination through approximately 28 days after study vaccination.
- 4. New onset chronic medical conditions (NOCMCs) and adverse events of special interest (AESI) NOCMC's will be assessed throughout the follow-up period, while medically attended wheezing events (an AESI) will be collected through Day 29 post-vaccination.

#### 4.5.2. Immunogenicity Variables

Humoral immune response will be assessed from venous blood samples collected at screening and on Days 1, 15, 29, and 181

Mucosal immune response will be determined by ELISA on specimens collected by nasal wick at screening for baseline immunology and again on Day 29 and Day 181.

Immunogenicity will be assessed by the Vanderbilt Vaccine Research Program Laboratory.

#### 4.5.3. Nasal Clearance Variables

Nasal clearance of *B. pertussis* will be determined by culture on specimens collected by nasal swab. The nasopharyngeal culture result will be reported as a binary outcome (i.e. bacteria detected / no bacteria detected) at Day 29 and Day 46 for subjects who remained positive at Day 29.

#### 5. SAMPLE SIZE CONSIDERATIONS

This study is planned to enroll approximately 50 healthy adults randomized into four treatment groups in a 3:3:3:1 ratio, as described in Section 4.4.3. Table 3 and Table 4 in the appendices describe the probability of observing safety events and the minimum detectable difference in seroconversion rates for the planned sample size.

Table 3 indicates the probability of observing one or more safety events (such as solicited local or systemic reactogenicity events, or an unsolicited non-serious AE of a particular type) for a treatment arm with the assumed event frequency and for the given sample size. For example, for any of the treatment arms with a sample size of 15 subjects, there is a 79.4% probability of detecting an AE that occurs at a frequency of 10%, and a 14% probability if the AE occurs at a rate of 1%.

One of the secondary outcome measures is the proportion of subjects that achieve seroconversion to individual pertussis antigens (PT, FHA, PRN, and FIM 2/3) by serum IgG or IgA ELISA at Days 15, 29 and 181 for humoral immune response. Table 4 shows the minimum detectable differences with 80% power between the proportion of subjects attaining seroconversion in the BPZE1 by VaxINator group versus Placebo using a two-sided Fisher's Exact test and alpha = 0.05.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

#### **6.1.** General Principles

Unless otherwise noted, all continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. In general, all data will be listed, sorted by treatment group and subject, and when appropriate by visit number within subject. All summary tables will be structured with a column for each treatment in the order (BPZE1 10<sup>7</sup> CFU administered via VaxINator, BPZE1 10<sup>9</sup> CFU administered via VaxINator, BPZE1 10<sup>9</sup> CFU administered via needleless tuberculin syringe, placebo administered via VaxINator) and will be annotated with the total population size relevant to that table/treatment, including any missing observations.

#### **6.2.** Timing of Analyses

- The preliminary safety and immunogenicity analysis will be performed when all safety, reactogenicity, immunogenicity and *B. pertussis* colonization data through Day 46 (or Day 29 if no subjects remain colonized with *B. pertussis* at Day 29) are available.
- The final analysis will be performed after all clinical, safety, and reactogenicity data through approximately 180 days after the study vaccination are available. Once the last subject completes the last visit, the final clinical database will be cleaned, monitored and locked. Unblinded analyses of safety, reactogenicity, colonization, and available immunogenicity data will then be performed by the SDCC and will be included in the CSR.

### 6.3. Analysis Populations

Summaries and analysis of safety data will be presented for the Safety Population. Summaries and analysis of immunogenicity data will be presented for the Immunogenicity Population. If there are major protocol deviations, a per-protocol (PP) analysis may also be performed. Summaries and analysis of nasal colonization data will be presented for the PP Population. A tabular listing of all subjects, visits, and observations excluded from the analysis populations will be provided in the CSR (Listing 4, Appendix 16.2.3).

#### **6.3.1.** Safety Population

The Safety Population will consist of all subjects who have received the study vaccine and for whom any data on safety are available. Subjects will be classified according to the treatment received. The primary safety analysis will be done on this population.

#### 6.3.2. Immunogenicity Population

The Immunogenicity Population will include all subjects who have received the study vaccination and contributed both pre-vaccination samples and either at least one post vaccination sample for humoral immunogenicity testing for which valid results were reported, or at least one post vaccination nasal sample for which valid results were reported. Subjects will be classified according to the treatment received.

#### 6.3.3. Per Protocol Population

The Per Protocol (PP) Population will include all subjects in the immunogenicity population, with the following exclusions:

- Data from all available visits for subjects found to be ineligible at baseline.
- Data from all visits subsequent to major protocol deviations, such as:
  - Receipt of non-study licensed live vaccine within 30 days before or after the study vaccination,
  - Receipt of non-study licensed inactivated vaccine within 14 days before or after the study vaccination.
  - Receipt of immunosuppressive therapy (e.g., corticosteroids) within 30 days before or after the study vaccination.
- Data from any visit that occurs substantially out of window. Whether a visit that occurs substantially out of window will be determined jointly by the principal investigator, the Sponsor, and the SDCC.

For analyses using the PP population, subjects will be grouped based on study vaccinations received.

### 6.4. Covariates and Subgroups

The protocol does not define any formal subgroup analyses, and the study is not adequately powered to perform subgroup analyses.

### 6.5. Missing Data

All attempts will be made to collect all data per protocol. As missing data are expected to be minimal, no imputation will be performed for missing values. Any data point that appears to be erroneous or inexplicable based on clinical judgment will be investigated as a possible outlier. If data points are identified as outliers, sensitivity analyses will be performed to examine the impact of including or excluding the outliers. Any substantive differences in these analyses will be reported.

### 6.6. Interim Analyses and Data Monitoring

Interim analyses would only be used to terminate this trial in the event that unanticipated safety events deemed to be of sufficient concern require such action by the sponsor. These interim assessments will not be made based on testing a formal statistical hypothesis; therefore, p-value adjustment will not be made to any analyses.

#### **6.6.1.** Interim Safety Review

An ISM and SMC will be convened by DMID to review study progress and participant, clinical, safety, and reactogenicity data. An interim safety review may include enrollment and demographic information, medical history, concomitant medications, physical assessments, clinical laboratory values, dosing compliance, solicited and unsolicited AE/SAEs, and *B. pertussis* colonization data. Additional data may be requested by the SMC, and interim statistical reports may be generated as deemed necessary and appropriate by DMID. The SMC may receive data in aggregate and presented by treatment arm, including expected and observed rates of the expected AEs. The SMC will review grouped data in the closed session only. The SMC will meet and review this data at scheduled time points or ad hoc as needed during this trial as defined in the SMC charter. As an outcome of each review/meeting, the SMC will make a recommendation as to the advisability of proceeding with study vaccinations (as applicable), and to continue, modify, or terminate this trial.

Additionally, this trial will be monitored to determine if any of the halting rules described in Section 9.5 of the protocol are met.

A preliminary report prepared with data through Day 46 (or Day 29 if no subjects remain colonized with *B. pertussis* at the Day 29 visit) will be prepared. This report will include analyses of safety and immunogenicity data.

#### 6.6.2. Interim Immunogenicity Review

A preliminary report of safety and immunogenicity and *B. pertussis* colonization data through Day 46 (or Day 29 if no subjects remain colonized with *B. pertussis* at the Day 29 visit) will be prepared. The analyses presented in this report will be released while subjects remain in the trial for long-term safety and immunogenicity follow-up and will be included in the final analysis of these data.

#### 6.7. Multicenter Studies

Not applicable. This study will take place at a single VTEU site.

### 6.8. Multiple Comparisons/Multiplicity

This study was not designed to test any specific null hypothesis, and as such no adjustments for multiple testing are planned.

#### 7. STUDY SUBJECTS

#### 7.1. Disposition of Subjects

Table 13 will present a summary of the reasons that subjects were screened but not enrolled.

The composition of analysis populations, including reasons for subject exclusion, by treatment arm, is presented in Table 11. A listing of subjects excluded from each analysis population will be presented in Listing 4.

The disposition of subjects in the study will be tabulated by treatment group (Table 10). The table shows the total number of subjects screened, enrolled, receiving study product, completing the Day 8 visit, completing the Day 15 reactogenicity period, completing the Day 29 blood draw, terminated from study follow-up, and the number who completed the study.

A flowchart showing the disposition of study subjects, adapted from the CONSORT Statement [15] will be included (Figure 2). This figure will present the number of subjects screened, enrolled, lost to follow-up, and analyzed, by treatment arm.

A listing of subjects who terminated from study follow-up and the reason will be included in Listing 1.

#### 7.2. Protocol Deviations

A summary of subject-specific protocol deviations will be presented by the deviation category, deviation type, and treatment group for all enrolled subjects (Table 5.) Deviations that are considered major deviations that will be reviewed for possible subject exclusion from the per protocol population include: deviations related to eligibility/enrollment, treatment administration schedule, follow-up visit schedule, and study product or specimen temperature excursions. All subject-specific protocol deviations and non-subject specific protocol deviations will be included in Appendix 3 as data listings (Listing 2 and Listing 3, respectively.)

#### 8. EFFICACY EVALUATION

This study was not designed to test a specific null hypothesis, rather the primary objectives included assessing the safety and tolerability of lyophilized BPZE1 vaccine.

#### 8.1. Secondary Immunogenicity Analysis

Summaries and analysis of immunogenicity data will be presented for the immunogenicity and PP populations by treatment group.

Immune responses in terms of toxin-specific serum IgG and IgA antibody titers (PT, FHA, PRN, FIM 2/3) will be summarized at each time point. Analyses will include the Geometric Mean Titers (GMTs) along with corresponding 95% confidence intervals (Table 17, Table 18, Table 19, and Table 20) and Geometric Mean Fold Rise (GMFR) (Table 21, Table 22, Table 23, and Table 24), as well as the proportion of subjects achieving seroconversion (defined as 2-fold increase over baseline of GMT) for each antigen (PT, FHA, PRN, and FIM 2/3) and the proportion of subjects that achieved seroconversion for ≥ 1 (Table 25 and Table 26) and ≥ 2 (Table 27 and Table 28) antigens (PT, FHA, PRN, and FIM 2/3.) Rates of seroconversion will be compared using Barnard's exact test. Reverse cumulative distributions (RCD) curves will also be presented for PT, FHA, PRN, and FIM 2/3 antibody titers. Plots for each assay will be generated with four panels (prevaccination, Day 15, Day 29, and Day 181), and separate curves within each panel for each treatment group, as shown in Figure 3, Figure 4, Figure 5, and Figure 6. Individual immunogenicity response data will also be presented (Listing 7 and Listing 8.)

Immune responses in terms of the ratio of toxin-specific (PT, FHA, PRN, FIM 2/3) nasal mucosal IgA antibody to total nasal mucosal IgA antibody will be summarized at each time point (Table 29 and Table 30.) Analyses will include the geometric mean titer ratios (GMTR) of antigen-specific IgA to total IgA and corresponding 95% confidence intervals, along with fold change of the GMTR from baseline. The proportion of subjects achieving seroconversion, defined as ≥2-fold rise of the GMTR from baseline, to each antigen (PT, FHA, PRN, and FIM 2/3) will be reported (Table 29 and Table 30) as well as the proportion of subjects that achieve seroconversion by nasal aspirate ELISA to one or more (Table 31 and Table 32) antigens (PT, FHA, PRN, and FIM 2/3) at either or both of Day 29 and Day 181. Rates of seroconversion will be compared using Barnard's exact test. Reverse cumulative distributions (RCD) curves will also be presented for mucosal PT, FHA, PRN, and FIM 2/3 antibody titers. Plots for each assay will be generated with three panels (prevaccination, Day 15, Day 29, and Day 181), and separate curves within each panel for each treatment group, as shown in Figure 7 and Figure 8. Individual immunogenicity response data will also be presented (Listing 9.)

Subjects will be tested for *B. pertussis* colonization by culture at Day 29 and, if positive, again at Day 46. The proportion of subjects with positive *B. pertussis* culture will be reported for the PP population at each time point with corresponding 95% confidence intervals (Table 33.) Individual nasal colonization data will also be presented (Listing 13.)

No formal hypothesis testing is planned.

#### 9. SAFETY EVALUATION

All summaries and analysis of safety data will be presented for the Safety Analysis Population. Safety summaries will be presented overall and by treatment group.

Listings will be sorted by treatment group, subject ID, parameter (if applicable), and visit.

Continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum and minimum. All categorical measures will be summarized by the frequency and percentages (based on the non-missing sample size) of observed levels. The denominator for the percentages may be based on the number of non-missing observations for an assessment or based on the number of subjects in a population. This will be described for each table.

### 9.1. Demographic and Other Baseline Characteristics

Summaries of age, sex, ethnicity, and race will be presented by treatment group and overall (Table 14 and Table 15.) Ethnicity is categorized as Hispanic or Latino, or not Hispanic and not Latino. In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the CRF as "No" to each racial option.

Individual subject listings (Appendix 3) will be presented for all demographics (Listing 5;) pre-existing medical conditions (Listing 6;) vital signs and oral temperature (Listing 16;) and concomitant medications (Listing 18.)

#### 9.1.1. Prior and Concurrent Medical Conditions

All current illnesses and pre-existing medical conditions will be MedDRA® coded using MedDRA dictionary version 21.0 or higher. Summaries of subjects' pre-existing medical conditions will be presented by treatment group (Table 16.) Individual subject listings will be presented for all medical conditions (Listing 6.)

#### 9.1.2. Prior and Concomitant Medications

During screening, medications and vaccines used up to 30 days prior will be solicited. Any medications used within 30 days prior to signing the informed consent form through 28 days after study vaccination (or early termination if prior to 28 days after study vaccination) will be recorded in the eCRFs. In addition, receipt of non-study vaccines will be solicited through approximately 28 days after study vaccination and recorded in the eCRFs.

Summaries of medications that were started prior to dosing and continuing at the time of dosing will be presented by WHO Drug Terms 2 and 3 and treatment group (Table 80.)

Individual subject listings will be presented for all concomitant medications (Listing 18.)

### **9.2.** Measurements of Treatment Compliance

Any subjects who are enrolled but not vaccinated will be presented by treatment group as part of the subject disposition table (Table 10.) Dates of treatment administration by treatment arm are presented in Table 12.)

#### 9.3. Adverse Events

When calculating the incidence of adverse events (i.e., on a per subject basis), each subject will only be counted once and any repetitions of adverse events within a subject will be ignored; the denominator will be

the total number of subjects in the safety population. All adverse events reported will be included in the summaries and analyses.

An overall summary of adverse events is presented in Table 34. Unsolicited adverse events occurring in more than 5% of subjects in any treatment group are presented in Table 35.

#### 9.3.1. Solicited Events and Symptoms

Systemic and mucosal (local) solicited adverse events will be collected from the time of study vaccination through 14 days after study vaccination. Systemic events include: fever, chills, fatigue, malaise, myalgia, arthralgia, headache, and hypersensitivity. Mucosal events include: runny nose, stuffy nose/congestion, nasal pain/irritation, epistaxis, sneezing, sinus pressure/pain, sore throat, cough, and shortness of breath. Solicited AEs will be summarized by severity for each day after the study vaccination (Days 1-14 post study vaccination) and as the maximum severity over all 15 days (Table 38, Table 40, Table 41, Table 42, Table 43, Table 44, Table 45, Table 46, Table 47, Table 48, Table 49, Figure 9, Figure 10, Figure 11, and Figure 12.) Severity will be graded on a scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). Grading scales for mucosal and systemic solicited adverse events are presented in Table 6, Table 7, and Table 8, respectively. Additionally, solicited AEs will be analyzed by taking the most severe response over the follow-up period, dichotomizing into a binary variable (none versus mild, moderate, or severe) and using standard techniques, such as exact confidence intervals, to summarize the proportion of subjects reporting each symptom, any local symptom, and any systemic symptom (Table 39.) Summaries of solicited AEs will be presented by treatment arm (Table 36.) The proportion of subjects reporting symptoms will be compared between treatment arms using Chi-square or Fisher's exact test (Table 37.) Solicited adverse events by subject will be presented in Listing 10 and Listing 11.

#### 9.3.2. Unsolicited Adverse Events

Unsolicited AEs will be coded by Medical Dictionary for Regulatory Activities (MedDRA) for preferred term and system organ class (SOC). Unsolicited SAEs will be collected from the time of study vaccination through approximately 6 months after study vaccination and reported by detailed listings showing the event description, MedDRA preferred term and SOC, relevant dates (study vaccinations and AEs), severity, relatedness, and outcome for each event (Listing 12). Non-serious unsolicited AEs will be collected from time of study vaccination through approximately 28 days after study vaccination and summarized as number and percentage of subjects reporting at least one event in each MedDRA preferred term and SOC, cross tabulated by severity and relationship to study product (Table 51, Table 52, Table 53, Table 54, Table 55, and Figure 13) and listed in Table 56. Additionally, the proportion of subjects and exact 95% confidence intervals of AEs in aggregate and by MedDRA categories will be computed (Table 50.)

### 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

The following listings will be presented including Subject ID, Adverse Event Description, Number of Days Post Dose (Duration), Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if not Related, and Outcome:

- Deaths and Serious Adverse Events (Table 56)
- Non-Serious Adverse Events (Table 57)
- New Onset Chronic Medical Conditions and Adverse Events of Special Interest (Table 58)

#### 9.5. Pregnancies

Safety population who become pregnant during the study, every attempt will be made to follow these subjects to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery. A listing of pregnancies and outcomes will be presented (Listing 19, Listing 20, Listing 21, Listing 22, and Listing 23.)

#### 9.6. Clinical Laboratory Evaluations

Clinical safety laboratory adverse events will be collected at the time of study vaccination through approximately 7 days after study vaccination (Day 8). Any clinical laboratory parameter that is abnormal at Day 8 will be repeated at the next study visit (or sooner if medically indicated) and followed until normal or stabilization. Parameters to be evaluated include white blood cell count, platelet count, hemoglobin concentration, alanine aminotransferase (ALT), and creatinine. Grading scales for safety laboratory parameters are presented in Table 9.

The number and percentage of subjects with at least one clinical safety laboratory abnormality through Day 8 is presented in the overall summary of adverse events (Table 34.)

The distribution of chemistry results by severity, time point, and treatment group will be presented in Table 61, Table 62, Table 63, Table 64, Table 65, Table 66, and Figure 14. The distribution of hematology results by severity, time point, and treatment group will be presented in Table 69, Table 70, Table 71, Table 72, Table 73, Table 74, Table 75, Table 76, and Figure 15. Descriptive statistics including mean, standard deviation, median, minimum and maximum values by time point, for each laboratory parameter, will be summarized in Table 67 and Table 68 (chemistry) and Table 77, Table 78, and Table 79 (hematology). Changes in laboratory values will be presented in Figure 16, Figure 17, Figure 18, Figure 19, and Figure 20.

Subject visits with abnormal laboratory results, Grade 1 severity or higher, will be presented in Table 59 and Table 60.

Listing 14 and Listing 15 will provide complete listings of individual clinical laboratory results with applicable reference ranges.

### 9.7. Vital Signs and Physical Evaluations

Vital sign measurements will include systolic blood pressure, diastolic blood pressure, oral temperature, and, pulse. Vital signs will be assessed at screening and at baseline prior to study vaccination. As abnormal vital signs are not expected, these will be listed by subject and time point (Listing 16.)

Full Physical Examinations will be performed at screening. Limited physical examinations focused on the nasopharynx, oropharynx, and lungs will be performed at Day 1, Day 8, and Day 15. If indicated based on review of interim medical history, a targeted physical examination will be performed at each in-clinic visit. A listing of physical exam findings will be presented (Listing 17.)

#### 9.8. Concomitant Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. A by-subject listing of concomitant medication use will be presented in Listing 18. The use of concomitant medications during the study will be summarized by ATC1, ATC2 code and treatment group for the Safety population (Table 80.)

### 9.9. Other Safety Measures

Not applicable.

### 10. PHARMACOKINETICS

Not applicable.

### 11. IMMUNOGENICITY

See Section 8.

### 12. OTHER ANALYSES

Not applicable.

#### 13. REPORTING CONVENTIONS

P-values ≥0.001 and ≤0.999 will be reported to 3 decimal places; p-values less than 0.001 will be reported as "<0.001" The mean, standard deviation, and other statistics will be reported to 1 decimal place greater than the original data. The minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as 2 decimal places; values greater than zero but <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values greater than zero but < 1% will be presented as "<1"; values greater than 99% but less than 100% will be reported as >99%. Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 significant figures.

### 14. TECHNICAL DETAILS

SAS version 9.4 or above will be used to generate all tables, figures and listings.

## 15. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

Not applicable.

#### 16. REFERENCES

- 1. Yeung, K.H.T., et al., An update of the global burden of pertussis in children younger than 5 years: a modelling study. Lancet Infect Dis, 2017. 17(9): p. 974-980.
- 2. Warfel, J.M., L.I. Zimmerman, and T.J. Merkel, Acellular pertussis vaccines protect against disease but fail to prevent infection and transmission in a nonhuman primate model. Proc Natl Acad Sci U S A, 2014. 111(2): p. 787-92.
- 3. Zhang, Q., et al., Prevalence of asymptomatic Bordetella pertussis and Bordetella parapertussis infections among school children in China as determined by pooled real-time PCR: a cross-sectional study. Scand J Infect Dis, 2014. 46(4): p. 280-7.
- 4. Ward, J.I., et al., Efficacy of an acellular pertussis vaccine among adolescents and adults. N Engl J Med, 2005. 353(15): p. 1555-63.
- 5. de Greeff, S.C., et al., Seroprevalence of pertussis in The Netherlands: evidence for increased circulation of Bordetella pertussis. PLoS One, 2010. 5(12): p. e14183.
- 6. Palazzo, R., et al., Evidence of increased circulation of Bordetella pertussis in the Italian adult population from seroprevalence data (2012-2013). J Med Microbiol, 2016.
- 7. Althouse, B.M. and S.V. Scarpino, Asymptomatic transmission and the resurgence of Bordetella pertussis. BMC Med, 2015. 13: p. 146.
- 8. Mielcarek, N., et al., Live attenuated B. pertussis as a single-dose nasal vaccine against whooping cough. PLoS Pathog, 2006. 2(7): p. e65.
- 9. Mielcarek, N., et al., Dose response of attenuated Bordetella pertussis BPZE1-induced protection in mice. Clin Vaccine Immunol, 2010. 17(3): p. 317-24.
- 10. Skerry, C.M., et al., A live attenuated Bordetella pertussis candidate vaccine does not cause disseminating infection in gamma interferon receptor knockout mice. Clin Vaccine Immunol, 2009. 16(9): p. 1344-51.
- 11. Feunou, P.F., et al., Genetic stability of the live attenuated Bordetella pertussis vaccine candidate BPZE1. Vaccine, 2008. 26(45): p. 5722-7.
- 12. Thorstensson, R., et al., A phase I clinical study of a live attenuated Bordetella pertussis vaccine-BPZE1; a single centre, double-blind, placebo-controlled, dose-escalating study of BPZE1 given intranasally to healthy adult male volunteers. PLoS One, 2014. 9(1): p. e83449.
- 13. Thorstensson, R., et al., A phase Ib (high dose), double-blind, single center, dose-escalating, placebocontrolled, randomized study of a live attenuated B. pertussis strain given as a single intranasal dose to healthy adult volunteers. 2017: on file at ILiAD Biotechnologies.
- 14. Locht, C., et al., Live attenuated pertussis vaccine BPZE1 protects baboons against B. pertussis disease and infection. J Infect Dis, 2017.
- 15. Drummond R. CONSORT Revised: Improving the Reporting of Randomized Clinical Trials. JAMA. 2001; 285(15):2006-2007.

### 17. LISTING OF TABLES, FIGURES, AND LISTINGS

Table, figure, and listing shells are presented in Appendix 1, Appendix 2, and Appendix 3, respectively. Please note that items marked with an asterisk (\*) are included in Preliminary Report.

### **APPENDICES**

### **APPENDIX 1. TABLE MOCK-UPS**

Tables that will be included in the Preliminary Report are indicated with an asterisk (\*) in the title.

### LIST OF TABLES

| Table 1: | Schedule of Study Procedures* | |
|---|---|---|
| Table 2: | Schedule of Study Procedures Secondary Table for Visits 4a and 4b*36 | |
| Table 3: | Probability (%) of Observing at Least One Adverse Event* | |
| Table 4: | Minimum Detectable Difference in Proportion of Subjects Attaining Seroconversion comparing Placebo versus the BPZE1 (10 <sup>7</sup> or 10 <sup>9</sup> CFU)* | |
| Table 5: | Distribution of Protocol Deviations by Category, Type, and Treatment Group38 | |
| Table 6: | Mucosal Reactogenicity Grading Scale* | |
| Table 7: | Subjective Systemic Reactogenicity Grading Scale* | |
| Table 8: | Quantitative Systemic Reactogenicity Grading Scale* | |
| Table 9: | Laboratory Adverse Event Grading Scale | |
| Table 10: | Subject Disposition by Treatment Group* | |
| Table 11: | Analysis Populations by Treatment Group* | |
| Table 12: | Dates of First Treatment by Treatment Group | |
| Table 13: | Ineligibility Summary of Screen Failures | |
| Table 14 | Summary of Categorical Demographic and Baseline Characteristics by Treatment Ground All Enrolled Subjects* | ıp, |
| Table 15: | Summary of Continuous Demographic and Baseline Characteristics by Treatment Groundle Subjects* | ıp, |
| Table 16: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Orga Class and Treatment Group | n |
| Table 17: | Serum IgA ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Interval by Time Point and Treatment Group, Immunogenicity Population*50 | |
| Table 18: | Serum IgA ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Interval by Time Point and Treatment Group, Per Protocol Population*51 | ıls |
| Table 19: | Serum IgG ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Interval by Time Point and Treatment Group, Immunogenicity Population*51 | ıls |
| Table 20: | Serum IgG ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Interval by Time Point and Treatment Group, Per Protocol Population*51 | ıls |
| Table 21: | Serum IgA ELISA Geometric Mean Fold Rise (GMFR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population*52 | |

### List of Tables (continued)

| Table 22: | Serum IgA ELISA Geometric Mean Fold Rise (GMFR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Per Protocol Population*56 |
|---|---|
| Table 23: | Serum IgG ELISA Geometric Mean Fold Rise (GMFR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population*56 |
| Table 24: | Serum IgG ELISA Geometric Mean Fold Rise (GMFR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Per Protocol Population*56 |
| Table 25: | Any One or More Serum Pertussis Antigens Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population* |
| Table 26: | Any One or More Serum Pertussis Antigens Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Per Protocol Population* |
| Table 27: | Any Two or More Serum Pertussis Antigens Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population*58 |
| Table 28: | Any Two or More Serum Pertussis Antigens Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Per Protocol Population* |
| Table 29: | Mucosal Ratio of PT-IgA to Total IgA ELISA Geometric Mean Titer Ratio (GMTR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population* |
| Table 30: | Mucosal IgA to Total IgA ELISA Geometric Mean Titer Ratio (GMTR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Per Protocol Population* |
| Table 31: | Any One or More Mucosal Pertussis Antigens Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population*63 |
| Table 32: | Any One or More Mucosal Pertussis Antigens Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Per Protocol Population*63 |
| Table 33: | Nasal Colonization Results by Time Point and Treatment Group, Per Protocol Population* |
| Table 34: | Overall Summary of Adverse Events* |
| Table 35: | Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety Population*67 |
| Table 36: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group* |
| Table 37: | Comparison of the Proportion of Subjects Experiencing Solicited Events by Treatment Group* |
| Table 38: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group* |
| Table 39: | Maximum Severity of Solicited Symptoms Dichotomized, by Symptom and Treatment Group |
# List of Tables (continued)

| Table 40: | Number and Percentage of Subjects Experiencing Systemic Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - BPZE1 10 <sup>7</sup> CFU by VaxINator * |
|---|---|
| Table 41: | Number and Percentage of Subjects Experiencing Systemic Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - BPZE1 10 <sup>9</sup> CFU by VaxINator * |
| Table 42: | Number and Percentage of Subjects Experiencing Systemic Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - BPZE1 10 <sup>9</sup> CFU by Syringe * |
| Table 43: | Number and Percentage of Subjects Experiencing Systemic Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - Placebo by VaxINator * |
| Table 44: | Number and Percentage of Subjects Experiencing Systemic Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - All Subjects *81 |
| Table 45: | Number and Percentage of Subjects Experiencing Local Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - BPZE1 10 <sup>7</sup> CFU by VaxINator *82 |
| Table 46: | Number and Percentage of Subjects Experiencing Local Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - BPZE1 109 CFU by VaxINator *84 |
| Table 47: | Number and Percentage of Subjects Experiencing Local Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - BPZE1 109 CFU by Syringe * .84 |
| Table 48: | Number and Percentage of Subjects Experiencing Local Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - Placebo by VaxINator *84 |
| Table 49: | Number and Percentage of Subjects Experiencing Local Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - All Subjects *84 |
| Table 50: | Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group* |
| Table 51: | Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group - BPZE1 10 <sup>7</sup> CFU by VaxINator*86 |
| Table 52: | Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group - BPZE1 10 <sup>9</sup> CFU by VaxINator* |
| Table 53: | Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group - BPZE1 10 <sup>9</sup> CFU by Syringe* |
| Table 54: | Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group – Placebo by VaxINator*.86 |
| Table 55: | Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group - All Subjects*86 |

# List of Tables (continued)

| Table 56: | Listing of Serious Adverse Events* |
|---|---|
| Table 57: | Listing of Unsolicited Non-Serious Adverse Events* |
| Table 58: | Listing of New Onset Chronic Medical Conditions and Adverse Events of Special Interest* |
| Table 59: | Listing of Abnormal Laboratory Results - Chemistry |
| Table 60: | Listing of Abnormal Laboratory Results - Hematology |
| Table 61: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter |
| Table 62: | Laboratory Results by Parameter Time Point, and Treatment Group – ALT95 |
| Table 63: | Laboratory Results by Parameter Time Point, and Treatment Group – Creatinine97 |
| Table 64: | Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter99 |
| Table 65: | Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – ALT |
| Table 66: | Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Creatinine |
| Table 67: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – ALT |
| Table 68: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Creatinine |
| Table 69: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Hematology Parameter |
| Table 70: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group - White Blood Cell Count |
| Table 71: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group — Platelet Count |
| Table 72: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group - Hemoglobin |
| Table 73: | Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Hematology Parameter115 |
| Table 74: | Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – White Blood Cell Count116 |
| Table 75: | Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Platelet Count |
| Table 76: | Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Hemoglobin |

# List of Tables (continued)

| Table 77: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – White Blood Cell Count |
|---|---|
| Table 78: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Platele Count |
| Table 79: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Hemoglobin |
| Table 80: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group |

### 9.5.1 Efficacy/Immunogenicity and Safety Measurements Assessed and Flow Chart

Table 1: Schedule of Study Procedures\*

| Study Visit Number | V00 | V01 | V02 | V03 | V04** | V05 | tion (if | f needed) |
|---|---|---|---|---|---|---|---|---|
| Study Day post study vaccination | Screening<br>(D-30 to D-1) | Enrollment<br>and Dose 1<br>D1 | D8±2d | D15±3d | D29±3d | D181±21d | Early Termination (if<br>needed) | Unscheduled (if needed) |
| Obtain Informed Consent∞ | X | $X^{\dagger}\neg$ | | | | | | |
| Collect Demographic Information | X | | | | | | | |
| Review Eligibility Criteria | X | $X^{\dagger}\neg$ | | | | | | |
| Medical History@ | X | $X^{\dagger}\neg$ | X | X | X | X | X | X |
| Concomitant Medications | $\mathbf{X}^{}$ | $X^{\sqrt{\uparrow} \neg}$ | X | X | x | | X (if prior to 28 days after study vaccination) | X (if prior to 28 days after<br>study vaccination) |
| Vital Signs <sup>\$</sup><br>(Oral Temperature <sup>%</sup> , Pulse, and BP) | X | $X^{\dagger}$ | | | | | X (may be obtained if indicated) | X (may be obtained if indicated) |
| Physical Examination! | X | $X^{\dagger 1}$ | $X^1$ | $X^1$ | (X) | (X) | (X) | (X) |
| Urine or Serum Pregnancy Test | Χ^ | Χ^ | | | | | | |
| Venous Blood Collection for Screening<br>Laboratory Assays <sup>2</sup> | X | | | | | | | |
| Venous Blood Collection for Safety<br>Laboratory Assays | | | X | | | | | |
| Venous Blood Collection for Serum<br>Antibody Assays | X | $X^{\dagger}$ | | X | X | x | $X^{\Omega}$ | |
| Venous Blood Collection for PBMC isolation and Future Research | | $X^{\dagger}$ | X | | X | X | $X^{\Omega}$ | |
| Nasal Sample Collection for Mucosal<br>Antibody Assays | X | | | | X | X | | |
| Nasal Sample Collection for <i>B. pertussis</i> Culture | | | | | X* | | | |
| Enrollment in AdvantageEDC <sup>SM</sup> and<br>Randomization | | $X^{\dagger}$ | | | | | | |

Table 1: Schedule of Study Procedures (continued)

| Study Visit Number | 000 | V01 | V02 | V03 | V04** | V05 | tion (if | f needed) |
|---|---|---|---|---|---|---|---|---|
| Study Day post study vaccination | Screening<br>(D-30 to D-1) | Enrollment<br>and Dose 1<br>D1 | D8±2d | D15±3d | D29±3d | D181±21d | Early Termination (if needed) | Unscheduled (if needed) |
| Pre-Administration Reactogenicity Assessments | | Χ <sup>†</sup> | | | | | | |
| Study Vaccination | | X | | | | | | |
| 2-hour Evaluation After Study Vaccination | | X | | | | | | |
| Post-Administration Reactogenicity Assessments | | X | | | | | X (if within 15 days after study vaccination) | X (if within 15 days after<br>study vaccination) |
| Distribute Memory Aid and Study-Related<br>Materials | | x | | | | | | |
| Review Memory Aid for Reactogenicity | | | X | X | | | X (if within 15 days after study vaccination) | X (if within 15 days after<br>study vaccination) |
| AE/SAE Assessment | | X& | X& | X& | X | X*** | X****(AEs if prior to 28 days after<br>study vaccination) | X*** (AEs if prior to 28 days after study vaccination) |

<sup>∞</sup> Prior to study procedures.

<sup>†</sup> Prior to study vaccination.

<sup>¬</sup> Review/confirm information or activity in subjects previously consented and screened.

<sup>@</sup> Complete medical history will be obtained by interview of the subjects at the screening visit and will be updated on Day 1 prior to study vaccination and interim medical history will be obtained by interview of the subjects at follow-up visits after study vaccination.

All concomitant medications taken, and vaccines received within 30 days prior to signing the informed consent and/or prior to study vaccination. Medications reported in the eCRF for this visit are limited to those taken within 30 days prior to signing the informed consent and/or prior to study vaccination.

<sup>\$</sup> Vital signs assessed on Day 1 prior to study vaccination will be considered as baseline.

<sup>%</sup> Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.

A physical examination will be performed by a study clinician licensed to make medical diagnoses and listed on the Form FDA 1572 as the site principal investigator or sub-investigator.

<sup>&</sup>lt;sup>1</sup> limited physical examination will be performed, focused on the nasopharynx, oropharynx, and lungs; in addition, a targeted physical examination will be performed, if indicated, based on review of interim medical history, by a study clinician.

<sup>()</sup> Targeted physical examination if indicated based on review of complete and any updates obtained by interview of subjects since the screening visit, by a study clinician licensed to make medical diagnoses and listed on the Form FDA 1572 as the site principal investigator or sub-investigator.

#### **Table 1: Schedule of Study Procedures** (continued)

- ^ Will be performed on all women of childbearing potential at screening and within 24 hours prior to study vaccination and results must be negative and known prior randomization and study vaccination.
- <sup>-</sup> PT and pertactin serum IgG
- & Inclusive of reactogenicity assessments performed on the day of study vaccination through 14 days after study vaccination.
- \*\*\* Assessment of AE/SAE limited to new-onset chronic medical conditions, AESI, and SAEs if after 28 days following the study vaccination.
- <sup>2</sup> To be performed locally by the site, and will include white blood cell count, hemoglobin, platelet count, alanine aminotransferase, serum creatinine, and HIV screening
- <sup>Ω</sup> Venous blood will only be obtained if the early termination visit occurs: 1) prior to Visit 2, 2) after day 14 post-vaccination but before Visit 3, or 3) at least 28 days following Visit 3.
- \*\* See Schedule of Events secondary table for Visits 4a and 4b.

Schedule of Study Procedures Secondary Table for Visits 4a and 4b\* Table 2:

| Study Visit Number | V4a** | V4b***<br>(Phone<br>call) |
|---|---|---|
| Study Day post study vaccination | D46±3d | Day 50<br>±3 days |
| Nasal Sample Collection for B. pertussis Culture and immunological assays | X | |
| Prescription of Azithromycin 500 mg by mouth once daily | | X |
| Interim Medical History | X | |
| SAE Assessment | X | |
| Targeted Physical Examination, if indicated | X | |

<sup>\*\*</sup>Study visit only if nasal sample is positive for *B. pertussis* at Day 29
\*\*\*Study visit only if nasal sample is positive for *B. pertussis* at Day 46

## 9.7.1 Sample Size

Table 3: Probability (%) of Observing at Least One Adverse Event\*

| Event<br>Frequency | N = 5 | N=15 |
|---------------------|-------|------|
| ≥0.01%<br>Rare | <0.1 | <0.1 |
| ≥0.1%<br>Uncommon | 0.5 | 1.5 |
| ≥1%<br>Common | 4.9 | 14.0 |
| ≥10%<br>Very Common | 41.0 | 79.4 |

Table 4: Minimum Detectable Difference in Proportion of Subjects Attaining Seroconversion comparing Placebo versus the BPZE1 (10<sup>7</sup> or 10<sup>9</sup> CFU)\*

| Placebo<br>by VaxINator | BPZE1 (10 <sup>7</sup> or 10 <sup>9</sup><br>CFU)<br>by VaxINator | Assumed Proportion of Subjects Attaining Seroconversion (Placebo) | Proportion<br>of Subjects<br>Attaining Seroconversion<br>(BPZE1) | Minimum Detectable Difference<br>(Treatment – Placebo) |
|---|---|---|---|---|
| | N=15 | 0.00 | 0.41 | 0.41 |
| | | 0.01 | 0.43 | 0.42 |
| N=15 | | 0.05 | 0.54 | 0.49 |
| | | 0.10 | 0.63 | 0.53 |
| | | 0.20 | 0.76 | 0.56 |

### **10.2** Protocol Deviations

Table 5: Distribution of Protocol Deviations by Category, Type, and Treatment Group

| | | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | | BPZE1 10 <sup>9</sup><br>CFU by<br>Syringe<br>(N=X) | | Placebo by<br>VaxINator<br>(N=X) | | All Subjects (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| Eligibility/enrollment | Any type | | | | | | | | | | |
| | Did not meet inclusion criterion | x | х | х | х | х | х | х | х | х | х |
| | Met exclusion criterion | | | | | | | | | | |
| | ICF not signed prior to study procedures | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Treatment administration schedule | Any type | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | |
| | Missed treatment administration | | | | | | | | | | |
| | Delayed treatment administration | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Follow-up visit schedule | Any type | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Protocol procedure/assessment | Any type | | | | | | | | | | |
| | Incorrect version of ICF signed | | | | | | | | | | |
| | Blood not collected | | | | | | | | | | |
| | Nasal mucus not collected | | | | | | | | | | |
| | Other specimen not collected | | | | | | | | | | |
| | Too few aliquots obtained | | | | | | | | | | |
| | Specimen result not obtained | | | | | | | | | | |
| | Required procedure not conducted | | | | | | | | | | |

Table 5: Distribution of Protocol Deviations by Category, Type, and Treatment Group (continued)

| | | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | | BPZE1 10 <sup>9</sup><br>CFU by<br>Syringe<br>(N=X) | | Placebo by<br>VaxINator<br>(N=X) | | All Subjects (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| | Required procedure done incorrectly | | | | | | | | | | |
| | Study product temperature excursion | | | | | | | | | | |
| | Specimen temperature excursion | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Treatment administration | Any type | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | |
| | Study product temperature excursion | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Blinding policy/procedure | Any type | | | | | | | | | | |
| | Treatment unblinded | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Note: N= Number | of subjects in the Safety Pop | ulation | ı | 1 | ı | | ı | • | ı | 1 | |

# 12.2.2 Displays of Adverse Events

**Table 6:** Mucosal Reactogenicity Grading Scale\*

| Local Reaction | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Runny nose | Noticeable but does not interfere with daily activity | Moderate discomfort that interferes with daily activity | Significant discomfort/prevents daily activity or seeks medical care |
| Stuffy nose/congestion | Noticeable but does not interfere with daily activity | Moderate discomfort that interferes with breathing from nose | Unable to breathe through nose or seeks medical care |
| Nasal nain/Irritation | | Moderate discomfort that interferes with daily activity | Significant discomfort that prevents daily activity or seeks medical care |
| Epistaxis Total duration of all episodes in a 24-hour period <30 minutes | | Total duration of all episodes in a 24-hour period >30 minutes | Any bleeding that required visit for medical encounter |
| Sneezing | Sneezing Noticeable but does not interfere with daily activity | | Significant discomfort; prevents daily activity |
| Sinus pressure/pain | Noticeable but does not interfere with daily activity | Moderate discomfort that interferes with daily activity | Significant discomfort that prevents daily activity or seeks medical care |
| Sore/irritated throat Noticeable but does not interfere with eating or drinking | | Moderate discomfort that interferes with eating or drinking | Significant discomfort that prevents eating or drinking or seeks medical care |
| Cough | Noticeable but does not interfere with daily activity or sleeping | Frequent cough that interferes with daily activity or sleeping | Prevents daily activity, prevents sleep, or seeks medical care |
| Shortness of breath/wheezing Noticeable but does not with daily activit | | Moderate discomfort that interferes with daily activity | Significant discomfort/ prevents<br>daily activity or seeks medical<br>encounter |

**Table 7:** Subjective Systemic Reactogenicity Grading Scale\*

| Systemic (Subjective) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Feverishness (Chills/Shivering/Sweating) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Fatigue (Tiredness) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Malaise (General Unwell Feeling) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Myalgia (Body Aches/Muscular Pain) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Arthralgia (Joint Pain) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Headache | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Rash/Hypersensitivity | Pruritus with or without rash | Localized urticaria | Generalized urticaria, anaphylaxis, or angioedema or localized urticaria that requires medical encounter. |

**Table 8:** Quantitative Systemic Reactogenicity Grading Scale\*

| Systemic (Quantitative) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Fever <sup>s</sup> - oral <sup>†</sup> | 38.0°C – 38.4°C | 38.5°C – 38.9°C | >38.9°C |
| | 100.4°F – 101.1°F | 101.2°F – 102.0°F | >102.0°F |

<sup>#</sup> Oral temperature assessed on Day 1 prior to the first study vaccination will be considered as baseline.

<sup>§</sup> A fever can be considered not related to the study product if an alternative etiology can be documented.

<sup>†</sup> Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature

# 12.4.1 Individual Laboratory Measurements and Abnormal Laboratory Values

 Table 9:
 Laboratory Adverse Event Grading Scale

| Hematology | Protocol<br>Range | Reference<br>Range | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|---|---|
| WBC 10 <sup>3</sup> /μL (Decrease) | ≥3.9 | 3.9 – 10.7 | 2.5 - 3.8 | 1.5 – 2.4 | <1.5 |
| WBC 10 <sup>3</sup> /μL (Increase) | ≥3.9 | 3.9 – 10.7 | 10.8 – 15.0 | 15.1 – 20.0 | >20.0 |
| Hemoglobin g/dL (Decrease, Male) | ≥13.0 | 13.0 – 18.1 | 11.0 – 12.9 | 9.5 – 10.9 | <9.5 |
| Hemoglobin g/dL (Decrease, Female) | ≥11.8 | 11.8 – 16.0 | 10.1 – 11.7 | 8.5 – 10.0 | <8.5 |
| Platelet count 10 <sup>3</sup> /μL (Decrease) | ≥135 | 135 – 371 | 125 – 134 | 100 – 124 | <100 |
| Platelet count 10 <sup>3</sup> /μL (Increase) | ≥135 | 135 – 371 | 372 – 550 | 551 – 750 | >750 |

| Chemistry | Protocol<br>Range | Reference<br>Range | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|---|---|
| ALT U/L (Increase, Female) | <45 | 0-44 | 45 – 100 | 101 – 200 | >200 |
| ALT U/L (Increase, Male) | <62 | 0-61 | 62 – 138 | 139 – 275 | >275 |
| Creatinine mg/dL (Increase, Female) | ≤1.11 | 0.57-1.11 | 1.12 – 1.60 | 1.61 – 2.00 | >2.00 or requires dialysis |
| Creatinine mg/dL (Increase, Male) | ≤1.25 | 0.72-1.25 | 1.26 – 1.70 | 1.71 – 2.00 | >2.00 or requires dialysis |

### 14.1 Description of Study Subjects

### 14.1.1 Disposition of Subjects

**Table 10:** Subject Disposition by Treatment Group\*

| Subject | BPZE1 10 <sup>7</sup> CFU by<br>VaxINator<br>(N=X) | | VaxI | BPZE1 10 <sup>9</sup> CFU by<br>VaxINator<br>(N=X) | | BPZE1 10° CFU by<br>Syringe<br>(N=X) | | bo by<br>Nator<br>=X) | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Disposition | n | % | n | % | n | % | n | % | n | % |
| Screened | | | | | | | | | x | |
| Enrolled/Randomized | х | 100 | х | 100 | х | 100 | х | 100 | x | 100 |
| Received Treatment | х | xx | х | xx | х | xx | х | xx | x | xx |
| Completed Day 8 Visit | х | xx | х | xx | х | xx | х | xx | x | xx |
| Completed Day 15<br>Reactogenicity Period | х | xx | х | xx | x | xx | Х | xx | x | xx |
| Completed Day 29 Blood Draw | х | xx | х | xx | х | xx | х | xx | x | xx |
| Early Termination <sup>a</sup> | х | xx | х | xx | х | XX | Х | xx | х | xx |
| Completed Follow-up<br>(Study Day 181) <sup>b</sup> | х | xx | х | xx | X | xx | Х | XX | Х | xx |

Note: N=Number of subjects enrolled

<sup>&</sup>lt;sup>a</sup> Refer to Listing 1 (Appendix section 16.2.1) for reasons subjects terminated early.

<sup>&</sup>lt;sup>b</sup> Refer to Listing 4 (Appendix section 16.2.3) for reasons subjects are excluded from the Analysis populations.

Table 11: Analysis Populations by Treatment Group\*

| | | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | | BPZE1 10 <sup>9</sup><br>CFU by<br>Syringe<br>(N=X) | | Placebo by<br>VaxINator<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Analysis Populations | Reason Subjects Excluded | % | n | % | n | % | n | % | n | % | n |
| Safety Population | Any Reason | X | XX | х | XX | х | XX | х | XX | х | XX |
| | [Reason 1, for example: Did not meet eligibility criteria] | | | | | | | | | | |
| | [Reason 2] | | | | | | | | | | |
| | [Reason 3] | | | | | | | | | | |
| | [Reason 4] | | | | | | | | | | |
| Immunogenicity Population | Any Reason | | | | | | | | | | |
| | [Reason 1] | | | | | | | | | | |
| | [Reason 2] | | | | | | | | | | |
| | [Reason 3] | | | | | | | | | | |
| | [Reason 4] | | | | | | | | | | |
| Per Protocol Population | Any Reason | | | | | | | | | | |
| | [Reason 1] | | | | | | | | | | |
| | [Reason 2] | | | | | | | | | | |
| | [Reason 3] | | | | | | | | | | |
| | [Reason 4] | | | | | | | | | | |
| Note: N=Number of subje | cts enrolled | | | | | • | | • | • | | |

**Table 12:** Dates of First Treatment by Treatment Group

| Dates of Dosing | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|
| Total (Entire period of enrollment) | | | | | |
| DDMMMYYYY-DDMMMYYYY | X | х | Х | X | X |
| Note: N= Number of subjects in the Safety Population | n | • | • | • | • |

Table 13: **Ineligibility Summary of Screen Failures** 

| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | n <sup>a</sup> | % b |
|---|---|---|---|
| Inclusion and Exclusion | Number of subjects failing any eligibility criterion | x | 100 |
| Inclusion | Any inclusion criterion | x | XX |
| | [inclusion criterion 1] | x | XX |
| | [inclusion criterion 2] | x | XX |
| | [inclusion criterion 3] | x | XX |
| Exclusion | Any exclusion criterion | x | XX |
| | [exclusion criterion 1] | x | XX |
| | [exclusion criterion 2] | x | XX |
| | [exclusion criterion 3] | x | XX |
| 03.5 1 1 1 | | | |

 <sup>&</sup>lt;sup>a</sup> More than one criterion may be marked per subject.
 <sup>b</sup> Denominator for percentages is the total number of screen failures.

# 14.1.2 Demographic Data by Study Group

Table 14 Summary of Categorical Demographic and Baseline Characteristics by Treatment Group, All Enrolled Subjects\*

| | | CFI<br>VaxI | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | | BPZE1 109<br>CFU by<br>Syringe<br>(N=X) | | Placebo by<br>VaxINator<br>(N=X) | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % | n | % | n | % | n | % |
| Sex | Male | x | xx | х | xx | х | xx | х | xx | x | xx |
| | Female | | | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | X | XX | х | xx | x | XX | х | xx | x | xx |
| | Hispanic or Latino | | | | | | | | | : | |
| | Not Reported | | | | | | | | | | |
| | Unknown | | | | | | | | | : | |
| Race | American Indian or Alaska Native | X | XX | х | XX | х | XX | х | XX | х | xx |
| | Asian | | | | | | | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | | | | | | | |
| | Black or African American | | | | | | | | | : | |
| | White | | | | | | | | | | |
| | Multi-Racial | | | | | | | | | : | |
| | Unknown | | | | | | | | | | |
| Note: N= | All subjects enrolled | l | 1 | ı | 1 | ı | ı | ı | 1 | ı | 1 |

Table 15: Summary of Continuous Demographic and Baseline Characteristics by Treatment Group, All Enrolled Subjects\*

| Variable | Statistic | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) | All Subjects (N=X) |
|---|---|---|---|---|---|---|
| Age (Years) | Mean | xx | XX | XX | XX | xx |
| | Standard Deviation | XX | XX | XX | XX | xx |
| | Median | X | X | X | X | X |
| | Minimum | X | X | X | X | x |
| | Maximum | X | X | X | X | X |
| Note: N=All s | subjects enrolled | • | 1 | • | | • |

#### 14.1.3 Prior and Concurrent Medical Conditions

Table 16: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group

| | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | | BPZE1 109<br>CFU by<br>Syringe<br>(N=X) | | Placebo by<br>VaxINator<br>(N=X) | | All Subjects (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class | n | % | n | % | n | % | n | % | n | % |
| Any SOC | х | xx | х | xx | х | xx | х | xx | х | XX |
| [SOC 1] | | | | | | | | | | |
| [SOC 2] | | | | | | | | | | |

Note: N= Number of subjects in the Safety Population; n = Number of subjects reporting medical history within the specified SOC. A subject is only counted once per SOC.

# 14.2 Efficacy/Immunogenicity Data

Table 17: Serum IgA ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point and Treatment Group, Immunogenicity Population\*

| Antigen | Time Point | Statistic | BPZE1<br>10 <sup>7</sup> CFU<br>by<br>VaxINator<br>(N=X) | BPZE1<br>10° CFU<br>by<br>VaxINator<br>(N=X) | BPZE1<br>10° CFU<br>by<br>Syringe<br>(N=X) | Placebo<br>by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|---|
| Pertussis Toxin (PT) | | | | | | |
| | Day 1 Pre-Vaccination | n | X | х | X | х |
| | | GMT | X.X | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| | Day 15 Post-Vaccination | n | X | Х | X | х |
| | | GMT | X.X | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| | Day 29 Post-Vaccination | n | X | х | X | х |
| | | GMT | X.X | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| | Day 181 Post-Vaccination | n | X | Х | X | х |
| | | GMT | X.X | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| Filamentous Hemagglutinin (FHA) | | | | | | |
| | Day 1 Pre-Vaccination | n | X | х | X | х |
| | | GMT | x.x | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| | Day 15 Post-Vaccination | n | X | х | X | Х |
| | | GMT | X.X | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| | Day 29 Post-Vaccination | n | X | х | X | х |
| | | GMT | x.x | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| | Day 181 Post-Vaccination | n | х | х | X | х |
| | | GMT | x.x | x x | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| Pertactin (PRN) | | | | | | |
| | Day 1 Pre-Vaccination | n | Х | Х | X | х |
| | | GMT | x.x | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| | Day 1 Pre-Vaccination | GMT | X.X | хх | хх | Х |

Table 17: Serum IgA ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point and Treatment Group, Immunogenicity Population (continued)

| Antigen | Time Point | Statistic | BPZE1<br>10 <sup>7</sup> CFU<br>by<br>VaxINator<br>(N=X) | BPZE1<br>10° CFU<br>by<br>VaxINator<br>(N=X) | BPZE1<br>10° CFU<br>by<br>Syringe<br>(N=X) | Placebo<br>by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|---|
| | Day 15 Post-Vaccination | n | X | х | х | х |
| | | GMT | X.X | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| | Day 29 Post-Vaccination | n | X | х | X | х |
| | | GMT | X.X | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| | Day 181 Post-Vaccination | n | X | Х | X | х |
| | | GMT | x.x | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| Fimbriae (FIM) | | | | | | |
| | Day 1 Pre-Vaccination | n | X | х | X | х |
| | | GMT | X.X | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| | Day 15 Post-Vaccination | n | X | х | X | х |
| | | GMT | X.X | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| | Day 29 Post-Vaccination | n | X | х | X | х |
| | | GMT | X.X | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |
| | Day 181 Post-Vaccination | n | X | X | X | х |
| | | GMT | X.X | хх | хх | хх |
| | | 95% CI | x x, x.x | x x, x x | x x, x x | x x, x.x |

Note: N=Number of subjects in the Immunogenicity Population n=Number of subjects with results available at time point

#### Tables with similar format:

Table 18: Serum IgA ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population\*

Table 19: Serum IgG ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point and Treatment Group, Immunogenicity Population\*

Table 20: Serum IgG ELISA Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population\*

<sup>\*</sup>Day 181 time point will not be presented in Preliminary Analysis

Table 21: Serum IgA ELISA Geometric Mean Fold Rise (GMFR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population\*

| Antigen | Time Point | Statistic | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10°<br>CFU by<br>VaxINator<br>(N=X) | BPZE1<br>10 <sup>9</sup> CFU<br>by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|---|
| Pertussis Toxin (PT) | | | | | | |
| | Day 15 Post-Vaccination | n | X | х | Х | х |
| | | GMFR <sup>a</sup> | x x | x.x | x.x | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | 2-Fold Rise <sup>b</sup> | x x | x.x | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | x x | x.x | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| | Day 29 Post-Vaccination | n | х | Х | X | х |
| | | GMFR <sup>a</sup> | x x | X.X | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | x.x | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | хх | x.x | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| | Day 181 Post-Vaccination | n | X | X | X | х |
| | | GMFR <sup>a</sup> | хх | x.x | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | X.X | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | хх | x.x | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| | Any Time Point | n | х | х | X | х |
| | | 2-Fold Rise <sup>b</sup> | хх | X.X | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | хх | x.x | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |

Table 21: Serum IgA ELISA Geometric Mean Fold Rise (GMFR) and Seroconversion (2-Fold rise) by Time Point and Treatment Group, Immunogenicity Population (continued)

| Antigen | Time Point | Statistic | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1<br>10 <sup>9</sup> CFU<br>by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|---|
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| Filamentous Hemagglutinin<br>(FHA) | | | | | | |
| | Day 15 Post-Vaccination | n | Х | Х | X | Х |
| | | GMFR <sup>a</sup> | x x | x.x | X.X | x x |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | 2-Fold Rise <sup>b</sup> | x x | x.x | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | x x | x.x | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| | Day 29 Post-Vaccination | n | X | X | X | х |
| | | GMFR <sup>a</sup> | хх | x.x | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | x.x | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | хх | X.X | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| | Day 181 Post-Vaccination | n | Х | Х | X | Х |
| | | GMFR <sup>a</sup> | хх | x.x | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | 2-Fold Rise <sup>b</sup> | x x | x.x | x.x | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | хх | x.x | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| | Any Time Point | n | X | X | Х | X |
| | | 2-Fold Rise <sup>b</sup> | хх | x.x | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | x x | x.x | N/A | N/A |

Table 21: Serum IgA ELISA Geometric Mean Fold Rise (GMFR) and Seroconversion (2-Fold rise) by Time Point and Treatment Group, Immunogenicity Population (continued)

| Antigen | Time Point | Statistic | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10°<br>CFU by<br>VaxINator<br>(N=X) | BPZE1<br>10° CFU<br>by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|---|
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| Pertactin (PRN) | | | | | | |
| | Day 15 Post-Vaccination | n | X | X | X | х |
| | | GMFR <sup>a</sup> | x x | X.X | x.x | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | X.X | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | хх | X.X | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| | Day 29 Post-Vaccination | n | X | X | X | х |
| | | GMFR <sup>a</sup> | хх | X.X | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | X.X | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | хх | X.X | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| | Day 181 Post-Vaccination | n | X | X | х | х |
| | | GMFR <sup>a</sup> | хх | X.X | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | 2-Fold Rise <sup>b</sup> | x x | X.X | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | хх | x.x | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| | Any Time Point | n | х | Х | x | х |
| | | 2-Fold Rise <sup>b</sup> | хх | X.X | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |

Table 21: Serum IgA ELISA Geometric Mean Fold Rise (GMFR) and Seroconversion (2-Fold rise) by Time Point and Treatment Group, Immunogenicity Population (continued)

| Antigen | Time Point | Statistic | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10°<br>CFU by<br>VaxINator<br>(N=X) | BPZE1<br>10 <sup>9</sup> CFU<br>by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|---|
| | | Difference <sup>c</sup> | x x | X.X | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| Fimbriae (FIM) | Day 15 Post-Vaccination | n | х | x | X | х |
| | | GMFR <sup>a</sup> | x x | X.X | x.x | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | X.X | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | хх | x.x | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| | Day 29 Post-Vaccination | n | X | X | X | х |
| | | GMFR <sup>a</sup> | x x | X.X | x.x | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | 2-Fold Rise <sup>b</sup> | x x | X.X | x.x | хх |
| | | Difference <sup>c</sup> | x x | X.X | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | Day 181 Post-Vaccination | n | х | Х | X | х |
| | | GMFR <sup>a</sup> | x x | x.x | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | 2-Fold Rise <sup>b</sup> | x x | X.X | X.X | хх |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| | | Difference <sup>c</sup> | хх | X.X | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |
| | Any Time Point | n | X | X | Х | X |
| | | 2-Fold Rise <sup>b</sup> | хх | X.X | x.x | ХX |
| | | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |

Table 21: Serum IgA ELISA Geometric Mean Fold Rise (GMFR) and Seroconversion (2-Fold rise) by Time Point and Treatment Group, Immunogenicity Population (continued)

| Antigen | Time Point | Statistic | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1<br>10° CFU<br>by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|---|
| | | Difference <sup>c</sup> | хх | x.x | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0.xx | N/A | N/A |

#### Tables with similar format:

- Table 22: Serum IgA ELISA Geometric Mean Fold Rise (GMFR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Per Protocol Population\*
- Table 23: Serum IgG ELISA Geometric Mean Fold Rise (GMFR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population\*
- Table 24: Serum IgG ELISA Geometric Mean Fold Rise (GMFR) and Seroconversion (2-Fold Rise)
  Results by Time Point and Treatment Group, Per Protocol Population\*

n=Number of subjects with results available at time point

<sup>&</sup>lt;sup>a</sup> GMFR represents the geometric mean fold rise in antibody titer compared to pre-dose 1.

<sup>&</sup>lt;sup>b</sup> 2-Fold Rise represents the percentage of subjects with at least a 2-Fold Rise in antibody compared to pre-dose 1.

c vs. placebo

<sup>&</sup>lt;sup>d</sup>Barnard's Exact test

<sup>\*</sup>Day 181 time point will not be presented in Preliminary Analysis

Table 25: Any One or More Serum Pertussis Antigens Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population\*

| Time Point | Statistic | BPZE1 10 <sup>7</sup> CFU<br>by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup> CFU<br>by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup> CFU<br>by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|
| Day 15 Post-Vaccination | n | х | х | х | Х |
| | 2-Fold Rise <sup>a</sup> | x x | x x | x x | X.X |
| | 95% CI | x x, x x | x.x, x x | x.x, x x | x.x, x x |
| | Difference <sup>b</sup> | x x | хх | N/A | N/A |
| | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | p-value <sup>c</sup> | 0 xx | 0 xx | N/A | N/A |
| Day 29 Post-Vaccination | n | х | x | x | X |
| | 2-Fold Rise <sup>a</sup> | x x | x x | x x | X.X |
| | 95% CI | x x, x x | x.x, x x | x.x, x x | x.x, x x |
| | Difference <sup>b</sup> | x x | хх | N/A | N/A |
| | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | p-value <sup>c</sup> | 0 xx | 0 xx | N/A | N/A |
| Day 181 Post-Vaccination | n | х | х | x | Х |
| | 2-Fold Rise <sup>a</sup> | x x | хх | x x | X.X |
| | 95% CI | x x, x x | x.x, x x | x.x, x x | x.x, x x |
| | Difference <sup>b</sup> | x x | хх | N/A | N/A |
| | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | p-value <sup>c</sup> | 0 xx | 0 xx | N/A | N/A |
| Any Time Point | n | х | X | х | Х |
| | 2-Fold Rise <sup>a</sup> | x x | x x | x x | X.X |
| | 95% CI | x x, x x | x.x, x x | x.x, x x | x.x, x x |
| | Difference <sup>b</sup> | x x | x x | N/A | N/A |
| | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | p-value <sup>c</sup> | 0 xx | 0 xx | N/A | N/A |

n=Number of subjects with results available at time point

<sup>&</sup>lt;sup>a</sup> 2-Fold Rise represents the percentage of subjects with at least a 2-Fold Rise in one or more antibodies compared to pre-dose 1.

<sup>&</sup>lt;sup>b</sup> vs. placebo

<sup>&</sup>lt;sup>c</sup>Barnard's Exact test

<sup>\*</sup>Day 181 time point will not be presented in Preliminary Analysis

#### Tables with similar format:

- Table 26: Any One or More Serum Pertussis Antigens Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Per Protocol Population\*
- Table 27: Any Two or More Serum Pertussis Antigens Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population\*
- Table 28: Any Two or More Serum Pertussis Antigens Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Per Protocol Population\*

Table 29: Mucosal Ratio of PT-IgA to Total IgA ELISA Geometric Mean Titer Ratio (GMTR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population\*

| Antigen | Time Point | Statistic | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 109<br>CFU by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|---|
| Pertussis Toxin (PT) | | | | | | |
| | Day 29 Post-Vaccination | n | X | х | х | X |
| | | GMTR <sup>a</sup> | хх | хх | X.X | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | хх | X.X | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | Difference <sup>c</sup> | хх | хх | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0 xx | N/A | N/A |
| | Day 181 Post-Vaccination | n | X | x | X | X |
| | | GMTR <sup>a</sup> | хх | хх | X.X | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | хх | X.X | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | Difference <sup>c</sup> | хх | хх | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0 xx | N/A | N/A |
| | Any Time Point | n | X | х | X | X |
| | | 2-Fold Rise <sup>b</sup> | хх | хх | X.X | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | Difference <sup>c</sup> | хх | хх | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0 xx | N/A | N/A |
| Filamentous Hemagglutinin (FHA) | | | | | | |
| | Day 29 Post-Vaccination | n | X | х | X | X |
| | | GMTR <sup>a</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | хх | X.X | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | Difference <sup>c</sup> | хх | хх | N/A | N/A |

Table 29: Mucosal Ratio of PT-IgA to Total IgA ELISA Geometric Mean Titer Ratio (GMTR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population (continued)

| Antigen | Time Point | Statistic | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|---|
| | | 95% CI of<br>Difference | x x, x x | x x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0 xx | N/A | N/A |
| | Day 181 Post-Vaccination | n | X | X | х | Х |
| | | GMTR <sup>a</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | Difference <sup>c</sup> | хх | хх | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0 xx | N/A | N/A |
| | Any Time Point | n | X | X | X | X |
| | | 2-Fold Rise <sup>b</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | Difference <sup>c</sup> | хх | хх | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0 xx | N/A | N/A |
| Pertactin (PRN) | | | | | | |
| | Day 29 Post-Vaccination | n | х | X | Х | X |
| | | GMTR <sup>a</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | Difference <sup>c</sup> | хх | хх | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0 xx | N/A | N/A |
| | Day 181 Post-Vaccination | n | X | X | х | X |
| | | GMTR <sup>a</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |

Table 29: Mucosal Ratio of PT-IgA to Total IgA ELISA Geometric Mean Titer Ratio (GMTR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population (continued)

| Antigen | Time Point | Statistic | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|---|
| | | Difference <sup>c</sup> | хх | хх | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0 xx | N/A | N/A |
| | Any Time Point | n | х | X | х | X |
| | | 2-Fold Rise <sup>b</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | Difference <sup>c</sup> | хх | хх | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0 xx | N/A | N/A |
| Fimbriae (FIM) | | | | | | |
| | Day 29 Post-Vaccination | n | х | X | Х | X |
| | | GMTR <sup>a</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | Difference <sup>c</sup> | хх | хх | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0 xx | N/A | N/A |
| | Day 181 Post-Vaccination | n | х | X | х | X |
| | | GMTR <sup>a</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | 2-Fold Rise <sup>b</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | Difference <sup>c</sup> | хх | хх | N/A | N/A |
| | | 95% CI of<br>Difference | x x, x x | x x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0 xx | N/A | N/A |
| | Any Time Point | n | х | х | х | X |
| | | 2-Fold Rise <sup>b</sup> | хх | хх | x.x | хх |
| | | 95% CI | x x, x x | x x, x x | x x, x.x | x.x, x x |
| | | Difference <sup>c</sup> | хх | хх | N/A | N/A |

Table 29: Mucosal Ratio of PT-IgA to Total IgA ELISA Geometric Mean Titer Ratio (GMTR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population (continued)

| Antigen | Time Point | Statistic | BPZE1 10 <sup>7</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup><br>CFU by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|---|
| | | 95% CI of<br>Difference | x x, x x | x x, x x | N/A | N/A |
| | | p-value <sup>d</sup> | 0 xx | 0 xx | N/A | N/A |

n=Number of subjects with results available at time point

#### Tables with similar format:

Table 30: Mucosal IgA to Total IgA ELISA Geometric Mean Titer Ratio (GMTR) and Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Per Protocol Population\*

<sup>&</sup>lt;sup>a</sup> GMTR represents the geometric mean titer ratio to total IgA

<sup>&</sup>lt;sup>b</sup> 2-Fold Rise represents the percentage of subjects with at least a 2-Fold Rise in antibody compared to pre-dose 1.

<sup>&</sup>lt;sup>c</sup> vs. placebo

<sup>&</sup>lt;sup>d</sup>Barnard's Exact test

<sup>\*</sup>Day 181 time point will not be presented in Preliminary Analysis

Table 31: Any One or More Mucosal Pertussis Antigens Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Immunogenicity Population\*

| Time Point | Statistic | BPZE1 10 <sup>7</sup> CFU<br>by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup> CFU<br>by<br>VaxINator<br>(N=X) | BPZE1 10° CFU<br>by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|
| Day 29 Post-Vaccination | N | x | X | x | x |
| | 2-Fold Rise <sup>a</sup> | x x | хх | хх | X.X |
| | 95% CI | x x, x x | x.x, x x | x.x, x x | x.x, x x |
| | Difference <sup>b</sup> | x x | хх | N/A | N/A |
| | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | p-value <sup>c</sup> | 0 xx | 0 xx | N/A | N/A |
| Day 181 Post-Vaccination | N | х | x | х | х |
| | 2-Fold Rise <sup>a</sup> | x x | хх | хх | X.X |
| | 95% CI | x x, x x | x.x, x x | x.x, x x | x.x, x x |
| | Difference <sup>b</sup> | хх | хх | N/A | N/A |
| | 95% CI of<br>Difference | x x, x x | x.x, x x | N/A | N/A |
| | p-value <sup>c</sup> | 0 xx | 0 xx | N/A | N/A |

Tables with similar format:

Table 32: Any One or More Mucosal Pertussis Antigens Seroconversion (2-Fold Rise) Results by Time Point and Treatment Group, Per Protocol Population\*

<sup>&</sup>lt;sup>a</sup> 2-Fold Rise represents the percentage of subjects with at least a 2-Fold Rise in one or more antibodies compared to pre-dose 1.

<sup>&</sup>lt;sup>b</sup> vs. placebo

<sup>&</sup>lt;sup>c</sup>Barnard's Exact test

<sup>\*</sup>Day 181 time point will not be presented in Preliminary Analysis

**Nasal Colonization Results by Time Point and Treatment Group, Per Protocol Population\* Table 33:** 

| | | BPZE1 10 <sup>7</sup> CFU by<br>VaxINator | BPZE1 10 <sup>9</sup> CFU by<br>VaxINator | BPZE1 10 <sup>9</sup> CFU by<br>Syringe | Placebo by<br>VaxINator |
|---|---|---|---|---|---|
| Time Point | Statistic | (N=X) | (N=X) | (N=X) | (N=X) |
| Day 29 Post-Vaccination | Subjects with detectable B. pertussis, n | X | x | X | х |
| | Proportion of subjects with detectable <i>B. pertussis</i> | XX | xx | xx | xx |
| | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| Day 46 Post-Vaccination | Subjects with detectable B. pertussis, n | X | х | X | х |
| | Proportion of subjects with detectable <i>B. pertussis</i> | XX | xx | XX | xx |
| | 95% CI | x x, x x | x.x, x x | x x, x.x | x x, x x |
| Note: N=Number of subjects | in the Per Protocol Population | _ I | ı | ı | 1 |

### 14.3 Safety Data

# 14.3.1 Displays of Adverse Events

Table 34: Overall Summary of Adverse Events\*

| | BPZE1 10 <sup>7</sup> CFU by<br>VaxINator<br>(N=X) | | BPZE1 10 <sup>9</sup> CFU by<br>VaxINator<br>(N=X) | | BPZE1 10° CFU by<br>Syringe<br>(N=X) | | Placebo by<br>VaxINator<br>(N=X) | | All Subjects (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | n | % | n | % | n | % | n | % | n | % |
| At least one local solicited adverse event | x | X | X | X | X | X | X | x | X | X |
| At least one systemic solicited adverse event | Х | Х | х | Х | х | х | х | х | X | Х |
| At least one unsolicited adverse event | X | X | х | x | x | x | x | x | X | Х |
| At least one unsolicited non-serious adverse event through Day 29 | X | X | х | x | х | х | X | X | X | х |
| At least one related unsolicited adverse event | x | X | X | X | X | X | X | X | X | Х |
| Mild (Grade 1) | X | х | X | X | X | X | х | X | X | X |
| Moderate (Grade 2) | x | X | х | Х | х | х | X | х | х | X |
| Severe (Grade 3) | х | х | х | х | х | х | х | х | х | X |
| Not yet assessed | | | | | | | | | | |
| At least one severe (Grade 3) unsolicited adverse event | X | X | x | х | x | x | x | x | X | X |
| Related | x | x | х | х | x | x | x | x | x | x |
| Unrelated | x | х | х | X | X | X | x | х | х | х |
**Table 34: Overall Summary of Adverse Events** (continued)

| | | 0 <sup>7</sup> CFU by<br>Nator<br>=X) | VaxI | 0° CFU by<br>Nator<br>=X) | Syr | 0 <sup>9</sup> CFU by<br>inge<br>=X) | VaxI | bo by<br>Nator<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | n % | | n | % | n | % | n | % | n | % |
| At least one serious adverse event <sup>b</sup> | X | X | X | X | X | X | X | X | X | X |
| At least one related, serious adverse event | X | X | X | X | X | X | X | X | X | X |
| At least one adverse event leading to early termination <sup>c</sup> | X | Х | X | х | х | х | Х | х | х | X |
| At least one medically attended adverse event | x | X | X | X | X | X | х | x | X | x |
| At least one new onset chronic medical condition | х | x | x | x | x | x | X | x | x | X |
| At least one potentially immune mediated medical condition | X | X | X | X | X | X | X | х | X | X |

N = Number of subjects in the Safety Population

a Subjects are counted once for each category regardless of the number of events.

b A listing of Serious Adverse Events is included in Table 56.

c As reported on the Adverse Event eCRF.

Table 35: Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety Population\*

| Preferred Term | MedDRA System<br>Organ Class | | E1 10 <sup>7</sup> C<br>vaxINato<br>(N=X) | | | E1 10 <sup>9</sup> C<br>VaxINato<br>(N=X) | | | E1 10 <sup>9</sup> C<br>Syringe<br>(N=X) | | | Placebo b<br>VaxINato<br>(N=X) | | A | ll Subjec<br>(N=X) | ts |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events |
| Serious Adverse Events | | | | | | | | | | | | | | | | |
| All | All | X | X | X | X | Х | X | X | X | X | X | X | X | X | X | X |
| PT1 | SOC1 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Etc. | Etc. | | | | | | | | | | | | | | | |
| Other (Non-serious) Adverse Events | | | | | | | | | | | | | | | | |
| All | All | X | X | X | X | х | X | X | Х | X | X | X | X | X | X | X |
| PT1 | SOC1 | Х | х | X | X | х | х | Х | х | Х | Х | х | Х | X | х | х |
| Etc. | Etc. | | | | | | | | | | | | | | | |

N = number of subjects in the Safety Population (number of subjects at risk).

n= number of subjects reporting event.

Events= total frequency of events reported.

# **14.3.1.1** Solicited Adverse Events

Table 36: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Group\*

| | | b<br>VaxI | 10 <sup>7</sup> CFU<br>y<br>Nator<br>=X) | | b | Nator | BP | ZE1<br>b<br>Syri<br>(N= | inge | | VaxI | bo by<br>Nator<br>=X) | P | All Subjec<br>(N=X) | ts |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Any Symptom | х | xx | x x, x x | X | XX | x.x, x x | x | xx | x x, x.x | Х | xx | x x, x.x | x | XX | x x, x.x |
| Any Systemic<br>Symptom | | | | | | | | | | | | | | | |
| Fever | | | | | | | | | | | | | | | |
| Feverishness | | | | | | | | | | | | | | | |
| Fatigue (tiredness) | | | | | | | | | | | | | | | |
| Malaise (general unwell feeling) | | | | | | | | | | | | | | | |
| Myalgia (body aches /muscular pain) | | | | | | | | | | | | | | | |
| Arthralgia (joint pain) | | | | | | | | | | | | | | | |
| Headache | | | | | | | | | | | | | | | |
| Rash / hypersensitivity | | | | | | | | | | | | | | | |
| Any Local Symptom | | | | | | | | | | | | | | | |
| Runny nose | | | | | | | | | | | | | | | |
| Stuffy nose/congestion | | | | | | | | | | | | | | | |
| Nasal pain/ Irritation | | | | | | | | | | | | | | | |
| Epistaxis | | | | | | | | | | | | | | | |
| Sneezing | | | | | | | | | | | | | | | |
| Sinus pressure/pain | | | | | | | | | | | | | | | |
| Sore/irritated throat | | | | | | | | | | | | | | | |
| Cough | | | | | | | | | | | | | | | |
| Shortness of breath/wheezing | | | | | | | | | | | | | | | |
| Note: N= Number of | subje | cts in | the Safety | y Pop | oulatio | on | | | | | | | | | |

Table 37: Comparison of the Proportion of Subjects Experiencing Solicited Events by Treatment Group\*

| Symptom | Statistic | BPZE1 10 <sup>7</sup> CFU<br>by<br>VaxINator<br>(N=X) | BPZE1 10° CFU<br>by<br>VaxINator<br>(N=X) | BPZE1 10 <sup>9</sup> CFU<br>by<br>Syringe<br>(N=X) | Placebo by<br>VaxINator<br>(N=X) |
|---|---|---|---|---|---|
| Any Symptom | Proportion | x.xx | x.xx | x.xx | x xx |
| | 95% CI (for proportion) | x xx, x.xx | x xx, x.xx | x xx, x.xx | x xx, x xx |
| | Difference <sup>a</sup> | x.xx | x.xx | N/A | N/A |
| | 95% CI (for difference) | x xx, x.xx | x xx, x.xx | N/A | N/A |
| [Symptom 1] | Proportion | x.xx | x.xx | x.xx | x xx |
| | 95% CI (for proportion) | x xx, x.xx | x xx, x.xx | x xx, x.xx | x xx, x xx |
| | Difference <sup>a</sup> | x.xx | x.xx | N/A | N/A |
| | 95% CI (for difference) | x xx, x.xx | x xx, x.xx | N/A | N/A |

Note: N = Number of subjects in the Safety Population who received at least one dose

<sup>&</sup>lt;sup>a</sup> vs. placebo

Table 38: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group\*

| | | BPZ | ZE1 10 <sup>7</sup> C<br>VaxINato<br>(N=X) | FU by<br>or | BPZ | ZE1 10 <sup>9</sup> C<br>VaxINato<br>(N=X) | or | BPZ | E1 10 <sup>9</sup> C<br>Syringe<br>(N=X) | | | Placebo l<br>VaxINat<br>(N=X) | or | A | All Subjec<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Any Symptom | None | X | XX | x.x, x x | X | XX | x x, x.x | X | XX | x.x, x x | X | XX | x x, x.x | X | XX | x x, x.x |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Systemic Symptoms | | | | | | | | | | | | | | | | |
| Any Systemic Symptom | None | X | XX | x.x, x x | Х | XX | x x, x.x | X | XX | x.x, x x | X | XX | x x, x.x | X | XX | x x, x.x |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Fever | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Fatigue (tiredness) | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |

Table 38: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group (continued)

| | | BPZ | ZE1 10 <sup>7</sup> C<br>VaxINato<br>(N=X) | FU by<br>or | BPZ | ZE1 10 <sup>9</sup> C<br>VaxINat<br>(N=X) | or | BPZ | ZE1 10 <sup>9</sup> C<br>Syringe<br>(N=X) | 9 | | Placebo l<br>VaxINato<br>(N=X) | or | F | All Subjec<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Malaise (general unwell feeling) | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Myalgia (body aches /muscular pain) | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Arthralgia (joint pain) | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Rash / hypersensitivity | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |

Table 38: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group (continued)

| | | BPZ | ZE1 10 <sup>7</sup> C<br>VaxINato<br>(N=X) | FU by<br>or | BPZ | ZE1 10 <sup>9</sup> C<br>VaxINat<br>(N=X) | or | BPZ | E1 10 <sup>9</sup> C<br>Syringe<br>(N=X) | e | | Placebo l<br>VaxINato<br>(N=X) | or | 1 | All Subjection (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| <b>Local Symptoms</b> | | | | • | | | | | | | | | | | | |
| Any Local Symptom | None | X | XX | x.x, x x | X | XX | x x, x.x | X | XX | x.x, x x | X | XX | x x, x.x | X | XX | x x, x.x |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Runny nose | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Stuffy nose/congestion | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Nasal pain/ Irritation | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Epistaxis | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |

Table 38: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group (continued)

| | | BPZ | ZE1 10 <sup>7</sup> Cl<br>VaxINato<br>(N=X) | FU by<br>or | | ZE1 10 <sup>9</sup> C<br>VaxINat<br>(N=X) | or | BPZ | XE1 10 <sup>9</sup> C<br>Syringe<br>(N=X) | | | Placebo b<br>VaxINato<br>(N=X) | oy<br>or | F | All Subjec<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Sneezing | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Sinus pressure/pain | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Sore/irritated throat | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Cough | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |
| Shortness of breath/wheezing | None | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | |

Note: N = Number of subjects in the Safety Population who received the specified dose. Severity is the maximum severity reported over all solicited symptoms post dosing for each subject.

Table 39: Maximum Severity of Solicited Symptoms Dichotomized, by Symptom and Treatment Group

| | | BPZ | E1 10 <sup>7</sup> C<br>VaxINat<br>(N=X) | or | BPZ | E1 10 <sup>9</sup> C<br>VaxINat<br>(N=X) | or | BPZ | E1 10 <sup>9</sup> C<br>Syringe<br>(N=X) | : | ] | Placebo l<br>VaxINat<br>(N=X) | or | A | All Subject | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Any Symptom | None | Х | xx | x.x, x x | х | XX | x x, x x | х | xx | x x, x x | Х | XX | x x, x x | X | XX | x x, x.x |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Systemic Symptoms | | | • | | | • | <b>.</b> | | · II | W. | | II. | | | | |
| Any Systemic Symptom | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Fever | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |

Table 39: Maximum Severity of Solicited Symptoms Dichotomized, by Symptom and Treatment Group (continued)

| | | BPZ | E1 10 <sup>7</sup> C<br>VaxINat<br>(N=X) | or | BPZ | E1 10 <sup>9</sup> C<br>VaxINato<br>(N=X) | FU by<br>or | BPZ | E1 10 <sup>9</sup> C<br>Syringe<br>(N=X) | - | ] | Placebo b<br>VaxINato<br>(N=X) | y<br>or | A | .ll Subjec<br>(N=X) | ts |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Fatigue (tiredness) | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Malaise (general unwell feeling) | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Myalgia (body aches /muscular pain) | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Arthralgia (joint pain) | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |

Table 39: Maximum Severity of Solicited Symptoms Dichotomized, by Symptom and Treatment Group (continued)

| | | | E1 10 <sup>7</sup> C<br>VaxINate<br>(N=X) | or | | E1 10 <sup>9</sup> C<br>VaxINato<br>(N=X) | | BPZ | E1 10 <sup>9</sup> C<br>Syringe<br>(N=X) | | ] | Placebo b<br>VaxINato<br>(N=X) | ey<br>or | A | .ll Subjec<br>(N=X) | ts |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Headache | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Rash / hypersensitivity | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Local Symptoms | | | ·I | | | | II. | • | | · I | • | 1. | | I. | | |
| Any Local Symptom | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Runny nose | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |

Table 39: Maximum Severity of Solicited Symptoms Dichotomized, by Symptom and Treatment Group (continued)

| | | BPZ | E1 10 <sup>7</sup> C<br>VaxINat<br>(N=X) | or | BPZ | E1 10 <sup>9</sup> C<br>VaxINato<br>(N=X) | FU by<br>or | BPZ | E1 10 <sup>9</sup> C<br>Syringe<br>(N=X) | | ] | Placebo b<br>VaxINato<br>(N=X) | y<br>or | A | .ll Subjec<br>(N=X) | ts |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Stuffy nose/congestion | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Nasal pain/ Irritation | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Epistaxis | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Sneezing | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |

Table 39: Maximum Severity of Solicited Symptoms Dichotomized, by Symptom and Treatment Group (continued)

| | | | E1 10 <sup>7</sup> C<br>VaxINate<br>(N=X) | or | BPZ | E1 10 <sup>9</sup> C<br>VaxINato<br>(N=X) | FU by<br>or | BPZ | E1 10 <sup>9</sup> C<br>Syringe<br>(N=X) | : | | Placebo b<br>VaxINato<br>(N=X) | | A | All Subjec<br>(N=X) | ets |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Sinus pressure/pain | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Sore/irritated throat | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Cough | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |
| Shortness of breath/wheezing | None | | | | | | | | | | | | | | | |
| | Mild or Worse | | | | | | | | | | | | | | | |
| | Moderate or<br>Worse | | | | | | | | | | | | | | | |
| | Severe or Worse | | | | | | | | | | | | | | | |

Note: N = Number of subjects in the Safety Population. Severity is the maximum severity reported over all solicited symptoms post dosing for each subject.

Table 40: Number and Percentage of Subjects Experiencing Systemic Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - BPZE1 10<sup>7</sup> CFU by VaxINator \*

| | | | Dose<br>=X) | | t-Dose<br>(=X) | | / 1-2<br>=X) | | 3-4<br>=X) | | 7 5-6<br>=X) | Day<br>(N= | 7-8<br>=X) | Day<br>(N= | 9-10<br>=X) | Day 1 | | | 13-14<br>=X) | | 15+<br>=X) | Any<br>Do | Post-<br>ose <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | n | % | n | % | n | % | n | % | n | % | n |
| Any Systemic Symptom | None | х | хх | х | x.x | х | хх | х | x.x | Х | хх | х | хх | х | хх | Х | хх | х | хх | х | хх | Х | хх |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Fever | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Fatigue (tiredness) | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |

Table 40: Number and Percentage of Subjects Experiencing Systemic Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - BPZE1 10<sup>7</sup> CFU by VaxINator (continued)

| | | | -Dose<br>=X) | | -Dose<br>=X) | | 1-2<br>=X) | | 3-4<br>=X) | | 7 <b>5-6</b><br>= <b>X</b> ) | | 7-8<br>=X) | | 9-10<br>=X) | | 11-12<br>=X) | | 13-14<br>=X) | Day<br>(N= | | Any<br>Do | Post-<br>ose <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | n | % | n | % | n | % | n | % | n | % | n |
| Malaise<br>(general unwell feeling) | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Myalgia (body aches / muscular pain) | None | | | | | | | | | | | | | | | | | | | | | | |
| - | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Arthralgia (joint pain) | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |

Table 40: Number and Percentage of Subjects Experiencing Systemic Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - BPZE1 10<sup>7</sup> CFU by VaxINator (continued)

| BPZE1 10 <sup>7</sup> CFU by V | VaxINator (N=X | X) | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Dose=X) | | -Dose<br>=X) | | 7 1-2<br>=X) | | 3-4<br>=X) | | 5-6<br>=X) | Day<br>(N= | 7-8<br>=X) | | 9-10<br>=X) | | 11-12<br>=X) | | 13-14<br>=X) | Day<br>(N= | | | Post-<br>ose <sup>a</sup> |
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | n | % | n | % | n | % | n | % | n | % | n |
| Rash / hypersensitivity | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |

Severity is the maximum severity reported post dosing for each subject for each day.

#### Tables with similar format:

- Table 41: Number and Percentage of Subjects Experiencing Systemic Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group BPZE1 109 CFU by VaxINator \*
- Table 42: Number and Percentage of Subjects Experiencing Systemic Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group BPZE1 109 CFU by Syringe \*
- Table 43: Number and Percentage of Subjects Experiencing Systemic Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group Placebo by VaxINator \*
- Table 44: Number and Percentage of Subjects Experiencing Systemic Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group All Subjects \*

<sup>&</sup>lt;sup>a</sup>Indicates how many subjects had "None", "Mild", "Moderate", "Severe", or "Not Reported" as the maximum severity for any day.

Table 45: Number and Percentage of Subjects Experiencing Local Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group - BPZE1 10<sup>7</sup> CFU by VaxINator \*

| BPZE1 10 <sup>7</sup> CFU by | | Pr | e-Dose<br>N=X) | | st-Dose<br>N=X) | Da<br>(N | ny 1-2<br>N=X) | Da<br>(I | ny 3-4<br>N=X) | Da<br>(N | y 5-6<br>N=X) | Da<br>(N | ny 7-8<br>N=X) | Da ( | ay 9-10<br>N=X) | Da ( | y 11-12<br>N=X) | Da ( | y 13-14<br>N=X) | Da<br>(N | y 15+<br>N=X) | Any Po | ost- Dose <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | n | % | n | % | n | % | n | % | n | % | n |
| Any Local Symptom | None | х | хх | Х | X.X | X | хх | X | хх | X | хх | Х | хх | X | хх | X | x.x | X | хх | X | хх | х | хх |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Runny nose | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Stuffy nose/congestion | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Nasal pain/irritation | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Epistaxis | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | Ì | | | | | | İ | | | | | | | | | | | | | |

Table 45: Number and Percentage of Subjects Experiencing Local Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group -- BPZE1 10<sup>7</sup> CFU by VaxINator (continued)

| BPZE1 10 <sup>7</sup> CFU by | vaxinator (N=X | | | 1 | | ı | | ı | | | | | | ı | | | | | | 1 | | 1 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | e-Dose<br>N=X) | | t-Dose<br>N=X) | Da<br>(N | y 1-2<br>N=X) | Da<br>(N | ny 3-4<br>N=X) | Da<br>(N | y 5-6<br>N=X) | Da<br>(N | y 7-8<br>N=X) | Da<br>(N | y 9-10<br>N=X) | Day<br>(I | y 11-12<br>N=X) | Day<br>(I | y 13-14<br>N=X) | Da<br>(N | y 15+<br>N=X) | Any Po | st- Dose <sup>a</sup> |
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | n | % | n | % | n | % | n | % | n | % | n |
| Sneezing | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Sinus pressure/pain | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Sore/irritated throat | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |
| Cough | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | 1 | | | | | | | | | | | | | | | | | | | | | |

Table 45: Number and Percentage of Subjects Experiencing Local Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group -- BPZE1 10<sup>7</sup> CFU by VaxINator (continued)

| BPZE1 10 <sup>7</sup> CFU by Va | xINator (N=X) | ) | | | | | | | | | | | | | | | | | | _ | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | e-Dose<br>N=X) | | st-Dose<br>N=X) | | ny 1-2<br>N=X) | | ay 3-4<br>N=X) | | ny 5-6<br>N=X) | | ny 7-8<br>N=X) | | y 9-10<br>N=X) | | y 11-12<br>N=X) | | y 13-14<br>N=X) | | y 15+<br>N=X) | Any Pos | st- Dose <sup>a</sup> |
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | n | % | n | % | n | % | n | % | n | % | n |
| Shortness of breath/wheezing | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | |

Severity is the maximum severity reported post dosing for each subject for each day.

#### Tables with Similar Format:

- Table 46: Number and Percentage of Subjects Experiencing Local Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group BPZE1 109 CFU by VaxINator \*
- Table 47: Number and Percentage of Subjects Experiencing Local Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group BPZE1 109 CFU by Syringe \*
- Table 48: Number and Percentage of Subjects Experiencing Local Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group Placebo by VaxINator \*
- Table 49: Number and Percentage of Subjects Experiencing Local Solicited Events by Symptom, Severity, Day Post Dosing, and Treatment Group All Subjects \*

<sup>&</sup>lt;sup>a</sup>Indicates how many subjects had "None", "Mild", "Moderate", "Severe", or "Not Reported" as the maximum severity for any day.

#### 14.3.1.2 Unsolicited Adverse Events

Table 50: Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group\*

| MedDRA<br>System | MedDRA | | Vax | 10 <sup>7</sup> CFU<br>INator<br>N=X) | by | | Va | 10 <sup>9</sup> CFU<br>xINator<br>N=X) | by | | S | 10 <sup>9</sup> CFU<br>vringe<br>N=X) | by | | Va | acebo by<br>xINator<br>(N=X) | | | | ubjects<br>N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Organ<br>Class | Preferred<br>Term | n | % | 95%<br>CI | Events | n | % | 95% CI | Events | n | % | 95%<br>CI | Events | n | % | 95%<br>CI | Events | n | % | 95%<br>CI | Events |
| Any SOC | Any PT | X | XX | xx, xx | x | X | XX | xx, xx | X | X | XX | xx, xx | x | X | XX | xx, xx | x | X | XX | xx, xx | х |
| [SOC 1] | Any PT | | | | | | | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | | | | | | | |

Note: N = number of subjects in the Safety Population who received the specified dose. This table presents number and percentage of subjects. A subject is only counted once per PT.

Table 51: Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group - BPZE1 10<sup>7</sup> CFU by VaxINator\*

| | | | B | PZE1 1 | | U by V<br>= X) | axINa | tor |
|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class | Preferred Term | Severity | Rel | ated | | ot<br>ated | To | otal |
| | | | n | % | n | % | n | % |
| Any SOC | Any PT | Any Severity | х | xx | Х | xx | Х | XX |
| | | Mild | х | XX | X | XX | X | XX |
| | | Moderate | х | XX | X | XX | X | XX |
| | | Severe | х | XX | X | XX | X | XX |
| SOC 1 | Any PT | Any Severity | х | xx | х | xx | X | XX |
| | | Mild | х | xx | х | xx | X | XX |
| | | Moderate | х | xx | х | xx | X | XX |
| | | Severe | х | xx | х | xx | X | XX |
| | PT 1 | Any Severity | х | xx | х | xx | X | XX |
| | | Mild | х | xx | х | xx | X | XX |
| | | Moderate | х | xx | Х | xx | Х | XX |
| | | Severe | Х | xx | Х | xx | Х | xx |
| Note: N = Number of subjects i | in the Safety Population. | • | | | | | | |

#### Tables with similar format:

- Table 52: Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group BPZE1 10<sup>9</sup> CFU by VaxINator\*
- Table 53: Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term,
  Maximum Severity, Relationship, and Treatment Group BPZE1 10<sup>9</sup> CFU by Syringe\*
- Table 54: Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group Placebo by VaxINator\*
- Table 55: Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group All Subjects\*

# 14.3.2 Listing of Deaths, Other Serious and Significant Adverse Events

# Table 56: Listing of Serious Adverse Events\*

| Adverse<br>Event | No. of Days<br>Post Dose<br>(Duration) | No. of Days Post Dose the Event Became Serious | Reason<br>Reported as<br>an SAE | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Gr | oup: , Subject II | D: , AE Number | : | | | | | | | | |
| | | T | _ | | T | _ | | Г | I | | |
| Comments: | | | | | | | | | | | |
| Commission. | | | | | | | | | | | |
| Treatment Gr | oup: , Subject II | D: , AE Number | : | | | | | | | | |
| Comments: | | | | | | | | | | | |

# Table 57: Listing of Unsolicited Non-Serious Adverse Events\*

| Adverse Event | No. of Days<br>Post Dose<br>(Duration) | Severity | Relationship to<br>Study<br>Treatment | If Not Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred Term |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | o: , Subject ID: , Al | E Number: | | | | | | | |
| Comments: | | | | | | | | | |
| Treatment Group | o: , Subject ID: , Al | E Number: | | | | | | | |
| Comments: | • | • | | | | • | | | |

# Table 58: Listing of New Onset Chronic Medical Conditions and Adverse Events of Special Interest\*

| Adverse Event | No. of Days Post<br>Dose | Duration of Event | Severity | MedDRA<br>System Organ<br>Class | AESI? | NOCMC? | Relationship | Outcome |
|---|---|---|---|---|---|---|---|---|
| Treatment Group: , | Subject ID: , AE Nu | mber: | | | | | | |
| Comments: | | | | | | | | |
| T | Called ID. AT No. | 1 | | | | | | |
| Treatment Group: , | Subject ID: , AE Nu | mber: | | | | | | |
| Comments: | | | | | | | | |

# 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, but this is a placeholder for the CSR)

# 14.3.4 Abnormal Laboratory Value Listings (by Subject)

# **Table 59:** Listing of Abnormal Laboratory Results - Chemistry

| Subject<br>ID | Treatment<br>Group | Sex | Age<br>(years) | Planned<br>Time Point | Actual<br>Study Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship to<br>Treatment | If Not Related,<br>Alternate<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued Due<br>to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|

# Table 60: Listing of Abnormal Laboratory Results - Hematology

| Subject<br>ID | Treatment<br>Group | Sex | Age<br>(years) | Planned<br>Time Point | Actual<br>Study Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship to<br>Treatment | If Not Related,<br>Alternate<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued Due<br>to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|

# 14.3.5 Displays of Laboratory Results

# 14.3.5.1 Chemistry Results

Table 61: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter

| Any Chemistry Parameter | | | N | one | | ild /<br>nde 1 | | erate/<br>ide 2 | | ere/<br>de 3 | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | x | x | xx | x | xx | x | xx | х | xx | х | XX |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | |

Table 61: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter (continued)

| Any Chemistry Parameter | | | No | one | | ild /<br>ide 1 | | erate/<br>ide 2 | Sev<br>Gra | | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | |
| N. T. (M. D. D. L. D. | All Subjects | | | 1 1: | | | 1 1 | | | | | 1 6 |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N=Number of subjects in the Safety Population

Table 62: Laboratory Results by Parameter Time Point, and Treatment Group – ALT

| | | | N | one | Gra | ild/<br>nde 1<br>ow) | Gra | ild/<br>nde 1<br>igh) | Gra | lerate/<br>ade 2<br>ow) | Gra | erate/<br>ide 2<br>igh) | Gra | rere/<br>ade 3<br>ow) | Gra | rere/<br>ide 3<br>igh) | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | х | х | XX | х | xx | х | xx | х | XX | х | xx | х | xx | х | xx | х | xx |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |

Table 62: Laboratory Results by Parameter, Time Point, and Treatment Group – ALT (continued)

| | | | No | one | Mi<br>Gra<br>(Lo | | Gra | ild/<br>de 1<br>igh) | Gra | erate/<br>ide 2<br>ow) | Gra | erate/<br>ide 2<br>igh) | Gra | ere/<br>de 3<br>ow) | Gra | rere/<br>ide 3<br>igh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post<br>Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population

**Table 63:** Laboratory Results by Parameter Time Point, and Treatment Group – Creatinine

| | | | No | one | Gra | ild/<br>ide 1<br>ow) | Gra | ild/<br>ide 1<br>igh) | Gra | erate/<br>ade 2<br>ow) | Gra | erate/<br>ide 2<br>igh) | Gra | vere/<br>nde 3<br>ow) | Gra | rere/<br>ide 3<br>igh) | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | х | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |

Table 63: Laboratory Results by Parameter, Time Point, and Treatment Group – Creatinine (continued)

| | | | No | one | Mi<br>Gra<br>(Lo | | Gra | ild/<br>de 1<br>igh) | Gra | erate/<br>ide 2<br>ow) | Gra | erate/<br>ide 2<br>igh) | Gra | ere/<br>de 3<br>ow) | Gra | rere/<br>ide 3<br>igh) | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post<br>Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population

Table 64: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter

| | | | | Tild/<br>rade 1 | Mod<br>Gra | lerate/<br>ade 2 | Sev<br>Gra | rere/<br>ide 3 |
|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % |
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | х | x | xx | x | xx | x | xx |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |

Table 64: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter (continued)

| | | | Mi<br>Gra | ild/<br>de 1 | Mode<br>Gra | | | rere/<br>ide 3 |
|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % |
| Max Severity Post Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity of abnormal laboratory results related to study treatment experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population

Table 65: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – ALT

| | | | | lild/<br>ade 1 | Mo<br>Gi | derate/<br>rade 2 | Sev<br>Gra | vere/<br>nde 3 |
|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % |
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | х | x | xx | x | xx | x | xx |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| _ | All Subjects | | | | | | | |
Table 65: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – ALT (continued)

| | | | | lild/<br>ade 1 | | erate/<br>ide 2 | Sev<br>Gra | ere/<br>de 3 |
|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % |
| Max Severity Post Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity of abnormal laboratory results related to study treatment experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population

Table 66: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Creatinine

| | | | | lild/<br>ade 1 | Mo<br>Gi | derate/<br>rade 2 | Sev<br>Gra | vere/<br>nde 3 |
|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % |
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | х | x | xx | x | xx | x | xx |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| _ | All Subjects | | | | | | | |

Table 66: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Creatinine (continued)

| | | | | lild/<br>ade 1 | | erate/<br>ide 2 | Sev<br>Gra | ere/<br>de 3 |
|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % |
| Max Severity Post Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity of abnormal laboratory results related to study treatment experienced by each subject at any time point post baseline, including unscheduled assessments. N= Number of subjects in the Safety Population

Table 67: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – ALT

| Time Point | Treatment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | X | xx x | xx x | xx x | xx x, xx x |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| | Placebo<br>by VaxINator | | | | | |
| | All Subjects | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| | Placebo<br>by VaxINator | | | | | |
| | All Subjects | | | | | |
| Day 8, Change from Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| | Placebo<br>by VaxINator | | | | | |
| | All Subjects | | | | | |

**Table 68: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Creatinine** 

| Time Point | Treatment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | x | XX X | xx x | xx x | xx x, xx x |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| | Placebo<br>by VaxINator | | | | | |
| | All Subjects | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| | Placebo<br>by VaxINator | | | | | |
| | All Subjects | | | | | |
| Day 8, Change from Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| | Placebo<br>by VaxINator | | | | | |
| | All Subjects | | | | | |
| Note: N= Number of subjects in the Safety Po | pulation | 1 | <u> </u> | | | |

## 14.3.5.2 Hematology Results

## Table 69: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Hematology Parameter

| Any Hematology Parameter | | | N | one | | ild /<br>nde 1 | | erate/<br>ide 2 | | vere/<br>ade 3 | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | X | X | xx | x | xx | x | xx | x | xx | x | xx |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | |

Table 69: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Hematology Parameter (continued)

| Any Hematology Parameter | | | No | one | Mi<br>Gra | | Mode<br>Gra | erate/<br>de 2 | Sev<br>Gra | | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | n % | | % | n | % | n | % | n | % |
| Max Severity Post Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | |

Table 70: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – White Blood Cell Count

| | | | No | one | Gra | ild/<br>nde 1<br>ow) | Gra | ild/<br>ide 1<br>igh) | Gra | erate/<br>ide 2<br>ow) | Gra | erate/<br>ide 2<br>igh) | Gra | rere/<br>ide 3<br>ow) | Gra | rere/<br>ide 3<br>igh) | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | x | х | XX | Х | xx | x | xx | x | xx | x | xx | x | xx | x | xx | x | xx |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |

Table 70: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – White Blood Cell Count (continued)

| | | | No | one | Gra | ild/<br>de 1<br>ow) | Gra | ild/<br>de 1<br>igh) | Gra | erate/<br>ide 2<br>ow) | Gra | erate/<br>ide 2<br>igh) | Gra | ere/<br>de 3<br>ow) | Gra | rere/<br>ide 3<br>igh) | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post<br>Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |

Table 71: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Platelet Count

| | | | No | one | Gra | ild/<br>nde 1<br>ow) | Gra | ild/<br>nde 1<br>igh) | Gra | erate/<br>nde 2<br>ow) | Gra | erate/<br>ide 2<br>igh) | Gra | rere/<br>ade 3<br>ow) | Gra | rere/<br>ide 3<br>igh) | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | х | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |

Table 71: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Platelet Count (continued)

| | | | No | one | Gra | ild/<br>de 1<br>ow) | Gra | ild/<br>de 1<br>igh) | Gra | erate/<br>ide 2<br>ow) | Gra | erate/<br>ide 2<br>igh) | Gra | ere/<br>de 3<br>ow) | | ere/<br>de 3<br>gh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post<br>Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | | | | | | | |

Table 72: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Hemoglobin

| | | | N | lone | | ild/<br>nde 1 | | erate/<br>ade 2 | | vere/<br>nde 3 | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | X | х | xx | х | xx | х | xx | х | xx | х | xx |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | |

Table 72: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Hemoglobin (continued)

| | | | N | one | Mi<br>Gra | ild/<br>de 1 | Mode<br>Gra | | | rere/<br>ide 3 | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post<br>Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | | | | | |
| | All Subjects | | | | | | | | | | | |

Table 73: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Hematology Parameter

| | | | Mild/<br>Grade 1 | | | derate/<br>rade 2 | | ere/<br>de 3 |
|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | х | х | xx | х | xx | х | xx |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |
| Max Severity Post Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity of abnormal laboratory results related to study treatment experienced by each subject at any time point post baseline, including unscheduled assessments. N = Number of subjects in the Safety Population

Table 74: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – White Blood Cell Count

| | | | Mild/<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | X | X | xx | х | XX | Х | xx |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |
| Max Severity Post Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |

Table 75: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Platelet Count

| | | | Mild/<br>Grade 1 | | | erate/<br>ide 2 | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | x | X | XX | х | xx | х | xx |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |
| Max Severity Post Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |

Table 76: Abnormal Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Treatment Group – Hemoglobin

| | | | Mild/<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | x | X | XX | х | XX | х | XX |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |
| Max Severity Post Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | | | |
| | Placebo<br>by VaxINator | | | | | | | |
| | All Subjects | | | | | | | |

Table 77: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – White Blood Cell Count

| Time Point | Treatment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | X | XX X | xx x | xx x | xx x, xx x |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| | Placebo<br>by VaxINator | | | | | |
| | All Subjects | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| | Placebo<br>by VaxINator | | | | | |
| | All Subjects | | | | | |
| Day 8, Change from Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| | Placebo<br>by VaxINator | | | | | |
| | All Subjects | | | | | |

**Table 78: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Platelet Count** 

| Time Point | Treatment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | х | xx x | xx x | xx x | xx x, xx x |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| | Placebo<br>by VaxINator | | | | | |
| | All Subjects | | | | | |
| Day 8 | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| | Placebo<br>by VaxINator | | | | | |
| | All Subjects | | | | | |
| Day 8, Change from Baseline | BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| | BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| | Placebo<br>by VaxINator | | | | | |
| | All Subjects | | | | | |

Table 79: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Hemoglobin

| Treatment Group | N | Mean | Standard Deviation | Median | Min, Max |
|---|---|---|---|---|---|
| BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | X | xx x | XX X | xx x | xx x, xx x |
| BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| Placebo<br>by VaxINator | | | | | |
| All Subjects | | | | | |
| BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | |
| BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| Placebo<br>by VaxINator | | | | | |
| All Subjects | | | | | |
| BPZE1 10 <sup>7</sup> CFU<br>by VaxINator | | | | | |
| BPZE1 10 <sup>9</sup> CFU<br>by VaxINator | | | | | |
| BPZE1 10 <sup>9</sup> CFU<br>by Syringe | | | | | |
| Placebo<br>by VaxINator | | | | | |
| | BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by Syringe Placebo by VaxINator All Subjects BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by Syringe Placebo by VaxINator All Subjects BPZE1 10° CFU by VaxINator All Subjects BPZE1 10° CFU by VaxINator BPZE1 10° CFU by Syringe Placebo | BPZE1 10 <sup>7</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by Syringe Placebo by VaxINator All Subjects BPZE1 10 <sup>7</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by Syringe Placebo by VaxINator All Subjects BPZE1 10 <sup>7</sup> CFU by Syringe Placebo by VaxINator All Subjects BPZE1 10 <sup>7</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by Syringe Placebo | BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by Syringe Placebo by VaxINator All Subjects BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by Syringe Placebo by VaxINator All Subjects BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by Syringe Placebo | BPZE1 10 <sup>7</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by Syringe Placebo by VaxINator All Subjects BPZE1 10 <sup>7</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by Syringe Placebo by VaxINator All Subjects BPZE1 10 <sup>7</sup> CFU by VaxINator BPZE1 10 <sup>7</sup> CFU by VaxINator BPZE1 10 <sup>7</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator BPZE1 10 <sup>9</sup> CFU by VaxINator | BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by Syringe Placebo by VaxINator All Subjects BPZE1 10° CFU by VaxINator All Subjects BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by VaxINator BPZE1 10° CFU by Syringe Placebo by VaxINator All Subjects BPZE1 10° CFU by VaxINator BPZE1 10° CFU by Syringe Placebo |

### 14.4 Summary of Concomitant Medications

Table 80: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group

| WHO Drug Code | WHO Drug Code | BPZE1 10 <sup>7</sup> CFU by<br>VaxINator<br>(N=X) | | BPZE1 10 <sup>9</sup> CFU by<br>VaxINator<br>(N=X) | | BPZE1 10 <sup>9</sup> CFU by<br>Syringe<br>(N=X) | | Placebo by<br>VaxINator<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Level 1, Anatomic Group | Level 2, Therapeutic Subgroup | n | % | n | % | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | X | XX | X | xx | X | xx | Х | xx | x | xx |
| [ATC Level 1 - 1] | Any [ATC 1 – 1] | | | | | | | | | | |
| | [ATC 2 - 1] | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | |
| [ATC Level 1 – 2] | [ATC 2 - 1] | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | |

N = Number of subjects in the Safety Population. n=Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

# APPENDIX 2. FIGURE MOCK-UPS

Figures that will be included in the Preliminary Report are indicated with an asterisk (\*) in the title.

## LIST OF FIGURES

| Figure 1 | Schematic of Study Design* |
|---|---|
| Figure 2: | CONSORT Flow Diagram |
| Figure 3: | Reverse Cumulative Distribution of Serum IgA Antibody Titers by Time Point and Treatment Group, Immunogenicity Population* |
| Figure 4: | Reverse Cumulative Distribution of Serum IgA Antibody Titers by Time Point and Treatment Group, Per Protocol Population* |
| Figure 5: | Reverse Cumulative Distribution of Serum IgG Antibody Titers by Time Point and Treatment Group, Immunogenicity Population* |
| Figure 6: | Reverse Cumulative Distribution of Serum IgG Antibody Titers by Time Point and Treatment Group, Per Protocol Population* |
| Figure 7: | Reverse Cumulative Distribution of Mucosal IgA Antibody Titers by Time Point and Treatment Group, Immunogenicity Population* |
| Figure 8: | Reverse Cumulative Distribution of Mucosal IgA Antibody Titers by Time Point and Treatment Group, Per Protocol Population* |
| Figure 9: | Maximum Severity of Solicited Systemic Events (by Symptom)*129 |
| Figure 10: | Maximum Severity of Solicited Local Events (by Symptom)* |
| Figure 11: | Maximum Severity of Solicited Systemic Symptoms per Subject by Days Post Treatment* |
| Figure 12: | Maximum Severity of Solicited Local Symptoms by Days Post Treatment*130 |
| Figure 13: | Number and Severity of All Adverse Events by MedDRA® System Organ Class*131 |
| Figure 14: | Clinical Laboratory Results by Severity – Hematology |
| Figure 15: | Clinical Laboratory Results by Severity – Chemistry |
| Figure 16: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – White Blood Cell Count |
| Figure 17: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Platelet Count |
| Figure 18: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Hemoglobin |
| Figure 19: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – ALT |

| Statistical | Analysis Plan - | DMID Protocol: | 17-0010 |
|-------------|-----------------|----------------|---------|
| Appendix | 2 – Figure Moc | k-ups | |

| List | of | <b>Figures</b> | (continued) |
|------|----|----------------|-------------|
|------|----|----------------|-------------|

### 9.1 Overall Study Design and Plan Description

Figure 1 Schematic of Study Design\*



### 10.1 Disposition of Subjects

Figure 2: CONSORT Flow Diagram



## 14.2.2 Efficacy/Immunogenicity Response Figures by Measure, Treatment/Vaccination, and Time Point

Figure 3: Reverse Cumulative Distribution of Serum IgA Antibody Titers by Time Point and Treatment Group, Immunogenicity Population\*

[Implementation Note: A sample figure is shown below. The legend order will be BPZE1 10<sup>7</sup> by VaxINator, BPZE1 10<sup>9</sup> by VaxINator, BPZE1 10<sup>9</sup> by VaxINator, BPZE1 10<sup>9</sup> by VaxINator.]



### Figures with similar format:

- Figure 4: Reverse Cumulative Distribution of Serum IgA Antibody Titers by Time Point and Treatment Group, Per Protocol Population\*
- Figure 5: Reverse Cumulative Distribution of Serum IgG Antibody Titers by Time Point and Treatment Group, Immunogenicity Population\*
- Figure 6: Reverse Cumulative Distribution of Serum IgG Antibody Titers by Time Point and Treatment Group, Per Protocol Population\*
- Figure 7: Reverse Cumulative Distribution of Mucosal IgA Antibody Titers by Time Point and Treatment Group, Immunogenicity
  - Population\*
- Figure 8: Reverse Cumulative Distribution of Mucosal IgA Antibody Titers by Time Point and Treatment Group, Per Protocol Population\*

#### 14.3.1.1 Solicited Adverse Events

### Figure 9: Maximum Severity of Solicited Systemic Events (by Symptom)\*

[Implementation Note: A sample figure is shown below. The following solicited events will be included: fever, feverishness, fatigue (tiredness), malaise (general unwell feeling), myalgia (body aches/muscular pain), arthralgia (joint pain), headache, rash/hypersensitivity and any systemic. The following five panels will be shown: BPZE1 10<sup>7</sup> by VaxINator, BPZE1 10<sup>9</sup> by VaxINator, BPZE1 10<sup>9</sup> by Syringe, Placebo by VaxINator and All Subjects.]



Figure with Similar Format:

Figure 10: Maximum Severity of Solicited Local Events (by Symptom)\*

[Implementation Note: The following solicited events will be included: runny nose, stuffy nose/congestion, nasal pain/irritation, epistaxis, sneezing, sinus pressure/pain, sore/irritated throat, cough and shortness of breath/wheezing and any local. The following five panels will be shown: BPZE1 10<sup>7</sup> by VaxINator, BPZE1 10<sup>9</sup> by VaxINator, BPZE1 10<sup>9</sup> by Syringe, Placebo by VaxINator and All Subjects.]

Figure 11: Maximum Severity of Solicited Systemic Symptoms per Subject by Days Post Treatment\*

[Implementation Note: A sample figure is shown below. The following timepoints will be presented; Post-vaccination, Days 1-2, Days 3-4, Days 5-6, Days 7-8, Days 9-10, Days 11-12, Days 13-14, and Days15+. The following five panels will be shown: BPZE1 10<sup>7</sup> by VaxINator, BPZE1 10<sup>9</sup> by VaxINator, BPZE1 10<sup>9</sup> by Syringe, Placebo by VaxINator and All Subjects.]



Figure with Similar Format:

Figure 12: Maximum Severity of Solicited Local Symptoms by Days Post Treatment\*

[Implementation Note: The following timepoints will be presented; Pre-vaccination, Post-vaccination, Days 1-2, Days 3-4, Days 5-6, Days 7-8, Days 9-10, Days 11-12, Days 13-14, and Days15+. The following five panels will be shown: BPZE1 10<sup>7</sup> by VaxINator, BPZE1 10<sup>9</sup> by VaxINator, BPZE1 10<sup>9</sup> by Syringe, Placebo by VaxINator and All Subjects.]

#### 14.3.1.2 Unsolicited Adverse Events

### Figure 13: Number and Severity of All Adverse Events by MedDRA® System Organ Class\*

[Implementation Note: A sample figure is shown below. This will include NOCMC's and AESI's. The following five panels will be shown: BPZE1 10<sup>7</sup> by VaxINator, BPZE1 10<sup>9</sup> by VaxINator, BPZE1 10<sup>9</sup> by Syringe, Placebo by VaxINator and All Subjects.]



### 14.3.5 Displays of Laboratory Results

### Figure 14: Clinical Laboratory Results by Severity – Hematology

[Implementation Note: A sample figure is shown below. White blood cell count increased/decreased, platelet count increased/decreased and hemoglobin decreased will be presented. The following five panels will be shown: BPZE1 10<sup>7</sup> by VaxINator, BPZE1 10<sup>9</sup> by VaxINator, BPZE1 10<sup>9</sup> by Syringe, Placebo by VaxINator and All Subjects.]



Figure 15: Clinical Laboratory Results by Severity – Chemistry

[Implementation Note: A sample figure is shown below. Only Creatinine and ALT will be presented. The following five panels will be shown: BPZE1 10<sup>7</sup> by VaxINator, BPZE1 10<sup>9</sup> by VaxINator, BPZE1 10<sup>9</sup> by Syringe, Placebo by VaxINator and All Subjects.]



Figure 16: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – White Blood Cell Count

[Implementation note: A sample figure is presented below. A scatter plot (dot plot) will be generated that displays each subject's change from baseline at Day 8 with the two treatment groups side by side. Overlaid on this plot will be the mean and standard deviation bars. Y-axis should be labeled "[Parameter] Change from Baseline ([units])"



Figures with similar format:

- Figure 17: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group Platelet Count
- Figure 18: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group Hemoglobin
- Figure 19: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group ALT
- Figure 20: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group Creatinine

# APPENDIX 3. LISTINGS MOCK-UPS

Listings are not included in the Preliminary Report.

## **LISTINGS**

| Listing 1: | 16.2.1 Early Terminations | .137 |
|---|---|---|
| Listing 2: | 16.2.2.1: Subject-Specific Protocol Deviations | .138 |
| Listing 3: | 16.2.2.2: Non-Subject-Specific Protocol Deviations | 139 |
| Listing 4: | 16.2.3: Subjects Excluded from Analysis Populations | 140 |
| Listing 5: | 16.2.4.1: Demographic Data | 141 |
| Listing 6: | 16.2.4.2: Pre-Existing and Concurrent Medical Conditions | 142 |
| Listing 7: | 16.2.6.1: Individual Immunogenicity Response Data – Serum IgA | 143 |
| Listing 8: | 16.2.6.2: Individual Immunogenicity Response Data – Serum IgG | 143 |
| Listing 9: | 16.2.6.3: Individual Immunogenicity Response Data – Mucosal IgA | 143 |
| Listing 10: | 16.2.7.1: Solicited Events – Systemic Symptoms | 144 |
| Listing 11: | 16.2.7.2: Solicited Events – Local Symptoms | 145 |
| Listing 12: | 16.2.7.3: Unsolicited Adverse Events | 146 |
| Listing 13: | 16.2.7.4: Individual Nasal Colonization Data | 147 |
| Listing 14: | 16.2.8.1: Clinical Laboratory Results – Chemistry | 148 |
| Listing 15: | 16.2.8.2: Clinical Laboratory Results – Hematology | 149 |
| Listing 16: | 16.2.9.1: Vital Signs | 150 |
| Listing 17: | 16.2.9.2: Physical Exam Findings | 151 |
| Listing 18: | 16.2.10: Concomitant Medications | 152 |
| Listing 19: | 16.2.11.1: Pregnancy Reports – Maternal Information | .153 |
| Listing 20: | 16.2.11.2: Pregnancy Reports – Gravida and Para | 153 |
| Listing 21: | 16.2.11.3: Pregnancy Reports – Live Birth Outcomes | 154 |
| Listing 22: | 16.2.11.4: Pregnancy Reports – Still Birth Outcomes | 154 |
| Listing 23: | 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes | 154 |

## 16.1.6 Listing of Subjects Receiving Investigational Product

(not included in SAP, but this is a placeholder for the CSR)

## 16.2 Database Listings by Subject

# **16.2.1 Discontinued Subjects**

## **Listing 1:** 16.2.1 Early Terminations

| Treatment Group | Subject ID | Reason for Early Termination | Study Day |
|-----------------|------------|------------------------------|-----------|
#### **16.2.2 Protocol Deviations**

# **Listing 2:** 16.2.2.1: Subject-Specific Protocol Deviations

| Treatment<br>Group | Subject ID | DV Number | Deviation | Deviation<br>Category | Study Day | Reason for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation Resulted<br>in Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|

**Listing 3:** 16.2.2.2: Non-Subject-Specific Protocol Deviations

| Start Date | Deviation | End Date | Reason for<br>Deviation | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|

## 16.2.3 Subjects Excluded from Analysis

## Listing 4: 16.2.3: Subjects Excluded from Analysis Populations

| Treatment Group | Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason Subject Excluded |
|---|---|---|---|---|---|
| | | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Day x] | | |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

# 16.2.4 Demographic Data

# Listing 5: 16.2.4.1: Demographic Data

| Treatment Group | Subject ID | Sex | Age at Enrollment (years) | Ethnicity | Race |
|---|---|---|---|---|---|

## Listing 6: 16.2.4.2: Pre-Existing and Concurrent Medical Conditions

| Treatment<br>Group | Subject ID | MH Number | Medical History Term | Condition Start Day | Condition End Day | MedDRA System Organ Class | MedDRA Preferred Term |
|---|---|---|---|---|---|---|---|

## 16.2.6 Individual Immunogenicity Response Data

Listing 7: 16.2.6.1: Individual Immunogenicity Response Data – Serum IgA

| | | | | PT An | tibody | FHA A | ntibody | PRN A | ntibody | FIM 2/3 | Antibody |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Subject ID | Planned<br>Time Point | Actual<br>Study Day | Titer | Fold-Rise | Titer | Fold-Rise | Titer | Fold-Rise | Titer | Fold-Rise |

Listings with similar format:

Listing 8: 16.2.6.2: Individual Immunogenicity Response Data – Serum IgG

Listing 9: 16.2.6.3: Individual Immunogenicity Response Data – Mucosal IgA

#### 16.2.7 Adverse Events

## **Listing 10:** 16.2.7.1: Solicited Events – Systemic Symptoms

| Treatment Group | Subject ID | Post Dose Day | Assessmenta | Symptom | Severity | Attributed to Alternate Etiology?b | Alternate Etiology |
|---|---|---|---|---|---|---|---|
| | | | MA | | | | |
| | | | Clinic | | | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

<sup>&</sup>lt;sup>b</sup> Grade 3 events only.

**Listing 11:** 16.2.7.2: Solicited Events – Local Symptoms

| Treatment Group | Subject ID | Post Dose Day | Assessment <sup>a</sup> | Symptom | Severity |
|---|---|---|---|---|---|
| | | | MA | | |
| | | | Clinic | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

Listing 12: 16.2.7.3: Unsolicited Adverse Events

| Adverse Event | No. of Days<br>Post Dose<br>(Duration) | Severity | SAE? | Relationship to Study<br>Treatment | In Not Related,<br>Alternative Etiology | Action Taken with<br>Study Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Group: , Subject ID: , AE Number: | | | | | | | | | | |
| Comments: | | | | | | | | | | |
| Treatment Grou | ıp: , Subject ID | : , AE Numl | ber: | | | | | | | |
| Comments: | Comments: | | | | | | | | | |
| Note: For addit | Note: For additional details about SAEs, see Table 56. | | | | | | | | | |

# Listing 13: 16.2.7.4: Individual Nasal Colonization Data

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | B. pertussis Positive? |
|---|---|---|---|---|

## 16.2.8 Individual Laboratory Measurements

# **Listing 14:** 16.2.8.1: Clinical Laboratory Results – Chemistry

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual<br>Study Day | Sex | Age (years) | Laboratory Parameter (Units) | Result (Severity<br>Grade) | Reference Range<br>Low | Reference Range<br>High |
|---|---|---|---|---|---|---|---|---|---|

## **Listing 15:** 16.2.8.2: Clinical Laboratory Results – Hematology

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual<br>Study<br>Day | Sex | Age<br>(years) | Laboratory Parameter<br>(Units) | Result (Severity<br>Grade) | Reference Range<br>Low | Reference Range<br>High |
|---|---|---|---|---|---|---|---|---|---|

## 16.2.9 Vital Signs and Physical Exam Findings

Listing 16: 16.2.9.1: Vital Signs

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual Study Day | Temperature<br>(°C) | Systolic Blood Pressure (mmHg) | Diastolic Blood Pressure<br>(mmHg) | Pulse<br>(beats/min) |
|---|---|---|---|---|---|---|---|

Listing 17: 16.2.9.2: Physical Exam Findings

| Treatment<br>Group | Subject ID | Planned<br>Time Point | Actual<br>Study Day | Body System | Abnormal Finding | Reported as an AE?<br>(AE Description; Number) | If Yes, Adverse Event |
|---|---|---|---|---|---|---|---|
| | | | | | | No | |
| | | | | | | Yes, Solicited | [Solicited AE] |
| | | | | | | Yes, Unsolicited | [Unsolicited AE Desc.;<br>Number] |

#### **16.2.10** Concomitant Medications

# **Listing 18:** 16.2.10: Concomitant Medications

| Treatment<br>Group | Subject ID | CM Number | Medication | Medication<br>Start Day | Medication<br>End Day | Indication | Taken for an AE? | If Yes,<br>Adverse<br>Event | Taken for a condition on<br>Medical History?<br>(MH Description; Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | No | | | |
| | | | | | | | Yes, Solicited | [Solicited AE] | | |
| | | | | | | | Yes,<br>Unsolicited | [Unsolicited<br>AE Desc.;<br>Number] | | |

### 16.2.11 Pregnancy Reports

### **Listing 19: 16.2.11.1: Pregnancy Reports – Maternal Information**

| Treatment<br>Group | Subject<br>ID | Pregnancy<br>Number | Study Day<br>Corresponding<br>to Estimated<br>Date of<br>Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco,<br>Alcohol, or<br>Drug Use<br>During<br>Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

### Listing 20: 16.2.11.2: Pregnancy Reports – Gravida and Para

| | | | Live Births | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>PB <sup>a</sup> | Very<br>Early<br>PB <sup>a</sup> | Early<br>PB <sup>a</sup> | Late<br>PB <sup>a</sup> | Early<br>TB <sup>b</sup> | Full<br>TB <sup>b</sup> | Late<br>TB <sup>b</sup> | Post<br>TB <sup>b</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly<br>with<br>Previous<br>Pregnancy? |

Note: Gravida includes the current pregnancy, para events do not.

a Preterm Birth

b Term Birth

## **Listing 21:** 16.2.11.3: Pregnancy Reports – Live Birth Outcomes

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month of<br>Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Congenital Anomalies are included in the Adverse Event listing.

### **Listing 22:** 16.2.11.4: Pregnancy Reports – Still Birth Outcomes

| Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress<br>During<br>Labor and<br>Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy, Etiology<br>for Still Birth<br>Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

## **Listing 23:** 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of Initial Report | Fetus Number | Pregnancy Outcome<br>(for this Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|